CLINICAL TRIAL: NCT05405166
Title: A Randomized, Phase 3, Open Label Study Evaluating Subcutaneous Versus Intravenous Administration of Isatuximab in Combination With Pomalidomide and Dexamethasone in Adult Patients With Relapsed and/or Refractory Multiple Myeloma (RRMM)
Brief Title: SC Versus IV Isatuximab in Combination With Pomalidomide and Dexamethasone in RRMM
Acronym: IRAKLIA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC15951; U1111-1261-5846 (Registry Identifier: ICTRP); 2023-508869-32 (Registry Identifier: CTIS); 2021-002485-41 (EudraCT Number)
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Plasma Cell Myeloma Recurrent
MeSH Terms: interventions — isatuximab; Dexamethasone; pomalidomide; montelukast; Acetaminophen; Diphenhydramine; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Isatuximab Subcutaneous (SC) (Experimental): Isatuximab dose will be administered SC weekly for 4 weeks during Cycle 1 (Days 1, 8, 15, and 22) and Day 1 and 15 of subsequent cycles. Each cycle will be 28 days in duration. Pomalidomide dose will be taken orally on Day 1 to Day 21 of each cycle at the time that is the most convenient for the participants prior to or after isatuximab administration, preferably at the same time every day. Dexamethasone will be taken orally on Day 1, 8, 15 and 22 (to be repeated every 28 days). Participants may receive other treatments as background treatment and/or rescue medication.
  Interventions: Drug: Isatuximab SC; Drug: Dexamethasone; Drug: Pomalidomide; Drug: Montelukast; Drug: Paracetamol / Acetaminophen; Drug: Diphenhydramine; Drug: Methylprednisolone
- Isatuximab Intravenous (IV) (Active Comparator): Isatuximab dose will be administered via IV infusion weekly for 4 weeks during Cycle 1 (Days 1, 8, 15, and 22) and Day 1 and 15 of subsequent cycles. Each cycle will be 28 days. Pomalidomide dose will be taken orally on Day 1 to Day 21 of each cycle at the time that is the most convenient for the participants prior to or after isatuximab administration, preferably at the same time every day. Dexamethasone will be taken orally on Day 1, 8, 15 and 22 (to be repeated every 28 days). Participants may receive other treatments as background treatment and/or rescue medication.
  Interventions: Drug: Isatuximab IV; Drug: Dexamethasone; Drug: Pomalidomide; Drug: Montelukast; Drug: Paracetamol / Acetaminophen; Drug: Diphenhydramine; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Isatuximab IV — Pharmaceutical form: Concentrate solution for IV infusion; Route of administration: Intravenous
  Other Names: SAR650984; SARCLISA®
  Arms: Isatuximab Intravenous (IV)
Drug: Isatuximab SC — Pharmaceutical form: Solution for subcutaneous administration; Route of administration: Subcutaneous (SC)
  Other Names: SAR650984
  Arms: Isatuximab Subcutaneous (SC)
Drug: Dexamethasone — Pharmaceutical form: Tablet; Route of administration: Oral
Drug: Pomalidomide — Pharmaceutical form: hard capsules; Route of administration: Oral
  Other Names: Pomalyst or equivalent
Drug: Dexamethasone — Pharmaceutical form: As per local commercial product; Route of administration: Oral; Auxiliary Medicinal Product (AxMP) i.e., background treatment; ATC code: H02AB02
Drug: Montelukast — Pharmaceutical form: As per local commercial product; Route of administration: Oral; AxMP i.e., background treatment; ATC code: R03DC03
Drug: Paracetamol / Acetaminophen — Pharmaceutical form: As per local commercial product; Route of administration: Oral; AxMP i.e., background treatment; ATC code: N02BE01
Drug: Diphenhydramine — Pharmaceutical form: As per local commercial product; Route of administration: As premedication- oral; for management of infusion reactions-IV (or oral equivalent); AxMP i.e., background treatment and rescue medication (in case of infusion reactions); ATC code: R06AA02
Drug: Methylprednisolone — Pharmaceutical form: As per local commercial product; Route of administration: As premedication-IV; for management of infusion reactions- IV (or oral equivalent); AxMP i.e., background treatment and rescue medication (in case of infusion reactions); ATC code: H02AB04

SUMMARY:
This is a randomized, multicenter, Phase 3, open-label study evaluating subcutaneous (SC) vs intravenous (IV) administration of isatuximab in combination with pomalidomide and dexamethasone (Pd) in RRMM patients (study participants) who have received at least 1 prior line of therapy including lenalidomide and a proteasome inhibitor (PI). Eligible participants will be randomized 1:1 into 1 of 2 study arms:

Arm SC: Isatuximab SC + Pd

Arm IV: Isatuximab IV + Pd

Participants will be allowed to continue therapy until disease progression, unacceptable adverse events (AEs), participant request to discontinue therapy or any other reason, whichever comes first.

DETAILED DESCRIPTION:
Two study arms will be treated in 4-week cycles until disease progression, unacceptable adverse events (AEs), participant request to discontinue therapy or any other reason, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Participants with multiple myeloma who have received at least one prior line of anti-myeloma therapy, which must include lenalidomide and a proteasome inhibitor given alone or in combination.
* Measurable serum M-protein (≥ 0.5 g/dL) and/or urine M-protein (≥ 200 mg/24 hours) and/or serum free light chain (FLC) assay (Involved FLC assay ≥10 mg/dL and abnormal serum FLC ratio (<0.26 or >1.65)).

Exclusion Criteria:

* Primary refractory multiple myeloma participants
* Participants with prior anti-CD38 treatment: (a) administered less than 9 months before randomization or, (b) intolerant to the anti-CD38 previously received
* Prior therapy with pomalidomide
* Participants with inadequate biological tests.
* Significant cardiac dysfunction
* Participants diagnosed or treated for another malignancy within 3 years prior to randomization with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, and in situ malignancy, or low risk prostate cancer after curative therapy
* Concomitant plasma cell leukemia
* Active primary amyloid light -chain amyloidosis
* Known acquired immunodeficiency syndrome (AIDS)-related illness or known human immunodeficiency virus (HIV) disease requiring antiviral treatment
* Know active Hepatitis A infection. Current active or chronic hepatitis B (HBV) or hepatitis C (HCV) infection. Participants with chronic HBV or HCV disease that is controlled under antiviral therapy are allowed.
* Women of childbearing potential or male participant with women of childbearing potential who do not agree to use highly effective method of birth control

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2027-03-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (146):
- United States (23):
  - Mohtaseb Cancer Center and Blood Disorders Site Number : 8400028, Bullhead City, Arizona
  - Arizona Oncology Associates, PC - HAL- Site Number : 8400015, Prescott Valley, Arizona
  - Rocky Mountain Cancer Centers, LLP- Site Number : 8400021, Aurora, Colorado
  - Mayo Clinic- Site Number : 8400008, Jacksonville, Florida
  - BRCR Medical Center Inc Site Number : 8400030, Plantation, Florida
  - Centre for Cancer and Blood Disorders- Site Number : 8400026, Bethesda, Maryland
  - Hattiesburg Clinic Site Number : 8400006, Hattiesburg, Mississippi
  - Comprehensive Cancer Centers of Nevada- Site Number : 8400019, Las Vegas, Nevada
  - Atlantic Health System Site Number : 8400005, Morristown, New Jersey
  - New York Oncology Hematology, P.C.- Site Number : 8400017, Albany, New York
  - Novant Health- Site Number : 8400014, Charlotte, North Carolina
  - Novant Health Forsyth Medical Center Site Number : 8400114, Winston-Salem, North Carolina
  - Gabrail Cancer Center Site Number : 8400027, Canton, Ohio
  - Oncology_Hematology Care Clinical Trials, LLC- Site Number : 8400016, Cincinnati, Ohio
  - Oncology Associates Of Oregon, P.C.- Site Number : 8400018, Eugene, Oregon
  - Spoknwrd Clinical Trials Inc. Site Number : 8400023, Easton, Pennsylvania
  - Gibbs Cancer Center-Spartanburg Medical Center- Site Number : 8400002, Spartanburg, South Carolina
  - Texas Oncology Baylor Sammons- Site Number : 8400022, Dallas, Texas
  - University of Texas Southwestern- Site Number : 8400024, Dallas, Texas
  - Lumi Research- Site Number : 8400029, Kingwood, Texas
  - Texas Oncology - San Antonio- Site Number : 8400020, San Antonio, Texas
  - George E. Wahlen Salt Lake City VA Medical Center- Site Number : 8400011, Salt Lake City, Utah
  - UW Cancer Center at ProHealth Care Site Number : 8400001, Waukesha, Wisconsin
- Argentina (10):
  - Investigational Site Number : 0320007, CABA, Buenos Aires
  - Investigational Site Number : 0320001, CABA, Buenos Aires
  - Investigational Site Number : 0320002, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Investigational Site Number : 0320006, La Plata, Buenos Aires
  - Investigational Site Number : 0320003, CABA, Buenos Aires F.D.
  - Investigational Site Number : 0320008, CABA, Buenos Aires F.D.
  - Investigational Site Number : 0320005, CABA, Buenos Aires F.D.
  - Investigational Site Number : 0320010, Córdoba, Córdoba Province
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320009, Mendoza
- Australia (7):
  - Investigational Site Number : 0360007, Liverpool, New South Wales
  - Investigational Site Number : 0360004, Waratah, New South Wales
  - Investigational Site Number : 0360003, Wollongong, New South Wales
  - Investigational Site Number : 0360008, Adelaide, South Australia
  - Investigational Site Number : 0360009, Fitzroy, Victoria
  - Investigational Site Number : 0360006, Melbourne, Victoria
  - Investigational Site Number : 0360001, Richmond, Victoria
- Brazil (6):
  - NOHC - Nucleo de Oncologia e Hematologia do Ceara- Site Number : 0760006, Fortaleza, Ceará
  - OC ONCOCLINICAS MULTIHEMO ILHA DO LEITE Site Number : 0760007, Recife, Pernambuco
  - CHN - Complexo Hospitalar de Niteroi Site Number : 0760008, Niterói, Rio de Janeiro
  - Hospital Mae de Deus Site Number : 0760003, Porto Alegre, Rio Grande do Sul
  - Clínica São Germano- Site Number : 0760001, São Paulo, São Paulo
  - Instituto COI de Educacao e Pesquisa- Site Number : 0760004, Rio de Janeiro
- Canada (3):
  - Investigational Site Number : 1240001, Toronto, Ontario
  - Investigational Site Number : 1240004, Greenfield Park, Quebec
  - Investigational Site Number : 1240003, Montreal, Quebec
- Chile (6):
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520006, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Viña del Mar, Región de Valparaíso
  - Investigational Site Number : 1520004, Santiago
  - Investigational Site Number : 1520001, Temuco
- China (15):
  - Investigational Site Number : 1560001, Beijing
  - Investigational Site Number : 1560022, Beijing
  - Investigational Site Number : 1560010, Changsha
  - Investigational Site Number : 1560006, Guangzhou
  - Investigational Site Number : 1560002, Hangzhou
  - Investigational Site Number : 1560020, Nanchang
  - Investigational Site Number : 1560019, Nanning
  - Investigational Site Number : 1560011, Qingdao
  - Investigational Site Number : 1560013, Shenyang
  - Investigational Site Number : 1560007, Tianjin
  - Investigational Site Number : 1560009, Tianjin
  - Investigational Site Number : 1560018, Tianjin
  - Investigational Site Number : 1560003, Wuhan
  - Investigational Site Number : 1560008, Wuhan
  - Investigational Site Number : 1560004, Zhengzhou
- Czechia (4):
  - Investigational Site Number : 2030005, Brno
  - Investigational Site Number : 2030003, Olomouc
  - Investigational Site Number : 2030006, Ostrava - Poruba
  - Investigational Site Number : 2030004, Prague
- France (7):
  - Investigational Site Number : 2500002, Nantes
  - Investigational Site Number : 2500005, Paris
  - Investigational Site Number : 2500008, Périgueux
  - Investigational Site Number : 2500001, Poitiers
  - Investigational Site Number : 2500009, Saint-Etienne
  - Investigational Site Number : 2500003, Toulouse
  - Investigational Site Number : 2500007, Tours
- Germany (5):
  - Investigational Site Number : 2760005, Dresden
  - Investigational Site Number : 2760001, Hamburg
  - Investigational Site Number : 2760003, Heidelberg
  - Investigational Site Number : 2760006, Lübeck
  - Investigational Site Number : 2760007, Nuremberg
- Greece (5):
  - Investigational Site Number : 3000002, Athens
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000005, Ioannina
  - Investigational Site Number : 3000003, Pátrai
  - Investigational Site Number : 3000004, Thessaloniki
- Hungary (6):
  - Investigational Site Number : 3480002, Budapest
  - Investigational Site Number : 3480004, Budapest
  - Investigational Site Number : 3480003, Kaposvár
  - Investigational Site Number : 3480008, Pécs
  - Investigational Site Number : 3480005, Székesfehérvár
  - Investigational Site Number : 3480006, Szombathely
- Italy (8):
  - Investigational Site Number : 3800001, Meldola, Forlì-Cesena
  - Investigational Site Number : 3800006, Rome, Roma
  - Investigational Site Number : 3800004, Ancona
  - Investigational Site Number : 3800002, Bologna
  - Investigational Site Number : 3800005, Brescia
  - Investigational Site Number : 3800007, Napoli
  - Investigational Site Number : 3800008, Palermo
  - Investigational Site Number : 3800003, Pavia
- Japan (12):
  - Investigational Site Number : 3920001, Nagoya, Aichi-ken
  - Investigational Site Number : 3920007, Kamogawa-shi, Chiba
  - Investigational Site Number : 3920005, Higashiibaraki-gun, Ibaraki
  - Investigational Site Number : 3920010, Shiwa-gun, Iwate
  - Investigational Site Number : 3920012, Kamakura-shi, Kanagawa
  - Investigational Site Number : 3920003, Kyoto, Kyoto
  - Investigational Site Number : 3920006, Natori-shi, Miyagi
  - Investigational Site Number : 3920002, Okayama, Okayama-ken
  - Investigational Site Number : 3920011, Osaka, Osaka
  - Investigational Site Number : 3920008, Sunto-gun, Shizuoka
  - Investigational Site Number : 3920004, Shibuya-ku, Tokyo
  - Investigational Site Number : 3920009, Yamagata
- Norway (2):
  - Investigational Site Number : 5780002, Ålesund
  - Investigational Site Number : 5780001, Oslo
- Poland (3):
  - Investigational Site Number : 6160005, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160004, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160001, Lublin
- Spain (7):
  - Investigational Site Number : 7240003, Santander, Cantabria
  - Investigational Site Number : 7240004, Badalona, Catalunya [Cataluña]
  - Investigational Site Number : 7240007, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240001, Pamplona, Navarre
  - Investigational Site Number : 7240005, Madrid
  - Investigational Site Number : 7240006, Murcia
  - Investigational Site Number : 7240002, Salamanca
- Sweden (2):
  - Investigational Site Number : 7520001, Borås
  - Investigational Site Number : 7520003, Stockholm
- Taiwan (3):
  - Investigational Site Number : 1580001, Kaohsiung City
  - Investigational Site Number : 1580005, Tainan
  - Investigational Site Number : 1580002, Taipei
- Turkey (Türkiye) (7):
  - Investigational Site Number : 7920007, Ankara
  - Investigational Site Number : 7920009, Ankara
  - Investigational Site Number : 7920004, Bornova
  - Investigational Site Number : 7920003, Istanbul
  - Investigational Site Number : 7920005, Istanbul
  - Investigational Site Number : 7920008, Istanbul
  - Investigational Site Number : 7920001, Istanbul
- United Kingdom (5):
  - Investigational Site Number : 8260002, Leicester, Leicestershire
  - Investigational Site Number : 8260005, London, London, City of
  - Investigational Site Number : 8260001, Norwich, Norfolk
  - Investigational Site Number : 8260004, Birmingham
  - Investigational Site Number : 8260003, Derby

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org.

REFERENCES:
- [Derived] Ailawadhi S, Spicka I, Spencer A, Lu J, Oriol A, Ling S, Schjesvold F, Berkovits A, Hus M, Li C, Dimopoulos MA, Rajnics P, Besisik SK, Hungria V, Custidiano MDR, Parmar G, Leleu X, Li F, Cerchione C, Gomez C, Ishida T, Mateos MV, Buck TT, LeBlanc R, Minarik J, Goldschmidt H, Zhang R, Semiond D, Suzan F, Stefanova-Urena M, Koch V, Moreau P. Isatuximab Subcutaneous by On-Body Injector Versus Isatuximab Intravenous Plus Pomalidomide and Dexamethasone in Relapsed/Refractory Multiple Myeloma: Phase III IRAKLIA Study. J Clin Oncol. 2025 Aug;43(22):2527-2537. doi: 10.1200/JCO-25-00744. Epub 2025 Jun 3. PMID 40459178
- See also: EFC15951 Relapsed/Refractory Multiple Myeloma USA website — https://www.sanofistudies.com/S2PX/
- See also: EFC15951 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25235&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 120 sites in 21 countries. A total of 637 participants were screened from 23-Jun-2022 to 13-May-2024, of which 106 were screen failures. Screen failures were mainly due to not meeting eligibility criteria.
Pre-assignment Details: A total of 531 participants were randomized in a 1:1 ratio to receive isatuximab (Isa) either via intravenous (IV) or subcutaneous (SC) route in combination with pomalidomide and dexamethasone (Pd). Interim results are presented up to primary completion date (PCD) of 06-Nov-2024. Reasons for study discontinuation at PCD are presented. Each cycle=28 days.
Groups:
- Isa-IV + Pd: Participants received isatuximab 10 milligrams/kilogram (mg/kg) IV infusion once weekly (QW) (i.e. on Days 1, 8, 15 and 22) in Cycle 1 (28 days) and then 10 mg/kg every 2 weeks (Q2W) (i.e. on Days 1 and 15) of each subsequent 28-day cycle along with pomalidomide 4 mg orally on Days 1 to 21 of each 28-day cycle and dexamethasone 40 mg (or 20 mg for participant >=75 years) orally on Days 1, 8, 15, and 22 of each cycle until disease progression, unacceptable adverse events (AEs), participant request to discontinue treatment, or any other reason, whichever came first.
- Isa-SC + Pd: Participants received isatuximab 1400 mg SC injection administered via an on-body delivery system (OBDS) which is an investigational device injector QW (i.e on Days 1, 8, 15 and 22) in Cycle 1 (28 days) and then 1400 mg Q2W (i.e. on Days 1 and 15) of each subsequent 28-day cycle along with pomalidomide 4 mg orally on Days 1 to 21 of each 28-day cycle and dexamethasone 40 mg (or 20 mg for participant >=75 years) orally on Days 1, 8, 15, and 22 of each cycle until disease progression, unacceptable AEs, participant request to discontinue treatment, or any other reason, whichever came first.
Period: Overall Study
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Started (Randomized) | 268 | 263
Randomized and Treated | 264 | 263
Completed | 0 | 0
Not Completed | 268 | 263
Not completed — Death | 49 | 50
Not completed — Withdrawal by Subject | 10 | 3
Not completed — Ongoing at the time of PCD | 209 | 210

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed for all randomized population.
Groups:
- Isa-IV + Pd: Participants received isatuximab 10 mg/kg IV infusion QW (i.e. on Days 1, 8, 15 and 22) in Cycle 1 (28 days) and then 10 mg/kg Q2W (i.e. on Days 1 and 15) of each subsequent 28-day cycle along with pomalidomide 4 mg orally on Days 1 to 21 of each 28-day cycle and dexamethasone 40 mg (or 20 mg for participant >=75 years) orally on Days 1, 8, 15, and 22 of each cycle until disease progression, unacceptable AEs, participant request to discontinue treatment, or any other reason, whichever came first.
- Isa-SC + Pd: Participants received isatuximab 1400 mg SC injection administered via an OBDS which is an investigational device injector QW (i.e on Days 1, 8, 15 and 22) in Cycle 1 (28 days) and then 1400 mg Q2W (i.e. on Days 1 and 15) of each subsequent 28-day cycle along with pomalidomide 4 mg orally on Days 1 to 21 of each 28-day cycle and dexamethasone 40 mg (or 20 mg for participant >=75 years) orally on Days 1, 8, 15, and 22 of each cycle until disease progression, unacceptable AEs, participant request to discontinue treatment, or any other reason, whichever came first.
- Total: Total of all reporting groups
Arm/Group | Isa-IV + Pd | Isa-SC + Pd | Total
Number analyzed (Participants) | 268 | 263 | 531
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.7) | 65.7 (9.4) | 65.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 126 | 238
  Male | 156 | 137 | 293
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 58 | 53 | 111
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 14 | 8 | 22
  White | 184 | 184 | 368
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR by independent review committee (IRC) using 2016 international myeloma working group (IMWG) criteria:Percentage of participants with complete response (CR),stringent CR (sCR),very good partial response (VGPR) & partial response (PR).CR:negative immunofixation on serum and urine,disappearance of any soft tissue plasmacytomas (STP),<5% plasma cells in bone marrow (BM) aspirates & a normal free light chain(FLC)ratio (0.26-1.65).sCR:CR plus no clonal cells in BM biopsy. VGPR:serum & urine M-protein detectable by immunofixation, not electrophoresis;>=90% reduction in serum M-protein plus urine M-protein level<100mg/24hour(h);>=90% decrease in sum of maximal perpendicular diameter (SPD) compared to baseline in STP;FLC only:>=90% decrease in difference between involved and uninvolved FLC levels.PR:>=50% reduction of serum M-protein and reduction in 24h urine M-protein by >=90% or to <200mg/24h.In addition to above, if present at baseline,>=50% reduction in size SPD of STPs also required.
Time Frame: From first dose of study medication administration (Day 1) up to PCD (06-Nov-2024), approximately 28 months
Population: The intent-to-treat (ITT) population included all randomized population (all participants who had given their informed consent and for whom there was confirmation of successful allocation of a randomization number by the interactive response technology [IRT]). Percentages are rounded off to the tenth decimal place.
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 268 | 263
percentage of participants | 70.5 [0.6467 to 0.7591] | 71.1 [0.6522 to 0.7651]
Statistical Analysis 1: Comparison: Isa-IV + Pd vs Isa-SC + Pd; Test type: Non-Inferiority — Non-inferiority was concluded if lower limit of relative risk 95% confidence interval (CI) was greater or equal to 0.839; p = 0.0006, Farrington-Manning; Relative risk = 1.008, 95% CI 2-sided [0.903 to 1.126] — Two-sided 95% CI estimated using Farrington-Manning method

2. Primary Outcome: Observed Concentration Before Dosing (Ctrough) of Isatuximab at Steady State
Description: Ctrough at steady state was the observed plasma concentration collected on pre-dose at Cycle 6 Day 1 (equivalent to prior to Cycle 6 Day 1) of isatuximab administration dose.
Time Frame: Pre-dose at Cycle 6 Day 1
Population: Per Protocol-Pharmacokinetic (PP-PK) population: all randomized participants who met following: at least 11 Isa dose from Cycle 1 Day 1 to Cycle 5 Day 15 (1 dose omission permitted at Cycle 1 only); Isa pre-dose plasma concentration results from PK samples on Cycle 6 Day 1 collected within PP defined time window with adequate documentation of dosing and sampling dates and times.
Measure: Mean (Standard Deviation); unit: microgram/milliliter (mcg/mL)
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 121 | 121
microgram/milliliter (mcg/mL) | 340 (169) | 499 (259)
Statistical Analysis 1: Comparison: Isa-IV + Pd vs Isa-SC + Pd; Test type: Non-Inferiority — Applied anti-log procedure to convert original scale. Non-inferiority was concluded if lower limit of ratio of geometric mean 90% CI was greater or equal to 0.80; Ratio of geometric mean = 1.532, 90% CI 2-sided [1.316 to 1.784]

3. Secondary Outcome: Very Good Partial Response or Better Rate
Description: VGPR or better rate by IRC using 2016 IMWG criteria: Percentage of participants with sCR, CR, and VGPR. CR: negative immunofixation on serum and urine, disappearance of any STP, <5% plasma cells in BM aspirates & normal FLC ratio (0.26-1.65). sCR: CR plus no clonal cells in BM biopsy. VGPR: serum and urine M-protein detectable by immunofixation, not electrophoresis;>=90% reduction in serum M-protein plus urine M-protein level<100mg/24h;>=90% decrease in SPD compared to baseline in STP; FLC only:>=90% decrease in difference between involved and uninvolved FLC levels. Percentages are rounded off to the tenth decimal place.
Time Frame: From first dose of study medication administration (Day 1) up to PCD (06-Nov-2024), approximately 28 months
Population: The ITT population included all randomized population.
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 268 | 263
percentage of participants | 45.9 | 46.4
Statistical Analysis 1: Comparison: Isa-IV + Pd vs Isa-SC + Pd; A hierarchical test procedure was used to control the Type I error. Testing was performed sequentially for first 4 secondary endpoints in the order they are presented only if both co-primary endpoints achieved non-inferiority and continued when the previous endpoint was statistically significant at 1-sided significance level of 0.025; Test type: Non-Inferiority — Non-inferiority was concluded if lower limit of relative risk 95% CI was greater or equal to 0.6312; p < 0.0001, Farrington-Manning; Relative risk = 1.011, 95% CI 2-sided [0.841 to 1.215] — Two-sided 95% CI estimated using Farrington-Manning method

4. Secondary Outcome: Ctrough of Isatuximab at 4 Weeks (CT4W)
Description: The CT4W was the observed plasma concentrations collected on pre-dose at Cycle 2 Day 1 (equivalent to prior to Cycle 2 Day 1) of isatuximab administration dose.
Time Frame: Pre-dose at Cycle 2 Day 1 (at 4 weeks)
Population: The CT4W-PK population: all randomized participants who met following: all 4 Isa doses for Cycle 1 administered; Isa pre-dose plasma concentration results from PK samples on Cycle 2 Day 1 collected within PP defined time window with adequate documentation of dosing and sampling dates and times.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 126 | 131
mcg/mL | 302 (117) | 421 (215)
Statistical Analysis 1: Comparison: Isa-IV + Pd vs Isa-SC + Pd; A hierarchical test procedure was used to control the Type I error. Testing was performed sequentially for first 4 secondary endpoints in the order they are presented only if both co-primary endpoints achieved non-inferiority and continued when the previous endpoint was statistically significant at 1-sided significance level of 0.05; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Ratio of geometric mean = 1.302, 90% CI 2-sided [1.158 to 1.465]

5. Secondary Outcome: Percentage of Participants With Infusion Reactions
Description: Infusion reactions were graded using National Cancer Institute-Common Terminology Criteria for AE (NCI-CTCAE) version (v)5.0 criteria: Grade 1: mild transient reaction; infusion interruption not indicated; intervention not indicated. Grade 2: moderate reaction; therapy or infusion interruption indicated but responds promptly to symptomatic treatment; prophylactic medications indicated for <=24 hours. Grade 3/4: severe or life-threatening reaction (Grade 3: prolonged [not rapidly responsive to symptomatic medication and/or brief interruption of infusion]; recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae. Grade 4: life-threatening consequences; urgent intervention indicated). Percentage of participants who observed AE of infusion reactions were collected through the electronic case report form (eCRF) as assessed by investigators. Percentages are rounded off to the tenth decimal place.
Time Frame: From first dose of study medication (Day 1) up to 30 days after the last dose of study medication, approximately 28 months
Population: The safety population included ITT participants who received at least 1 dose or a part of a dose of the study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 264 | 263
percentage of participants | 25.0 [19.89 to 30.68] | 1.5 [0.42 to 3.85]
Statistical Analysis 1: Comparison: Isa-IV + Pd vs Isa-SC + Pd; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Fisher Exact; Relative risk = 0.061, 95% CI 2-sided [0.022 to 0.164] — Two-sided 95% CI estimated using Wald method

6. Secondary Outcome: Percentage of Participants Who Responded Very Satisfied and Satisfied to the 'Patient Experience and Satisfaction Questionnaire (PESQ-FU)': Satisfaction With Injection Method' (Item-8) at Cycle 5 Day 15
Description: The PESQ-FU consisting of 9 items has been designed to follow up on participant experience and satisfaction regarding the injection method (discomfort, pain, side effects, time saving and satisfaction) and study medication (side effects, worth taking, satisfaction and recommendation). This questionnaire has been adapted based on qualitative interviews with oncology participants. The responses to 'satisfaction with injection method' were recorded as 'very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied and very dissatisfied' at specified timepoints. The total percentage of participants who were very satisfied and satisfied with the injection method (item-8) at Cycle 5 Day 15 is reported here. Percentages are rounded off to the tenth decimal place.
Time Frame: Cycle 5 Day 15
Population: The ITT population included all randomized population.
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 268 | 263
percentage of participants | 53.4 | 70.0
Statistical Analysis 1: Comparison: Isa-IV + Pd vs Isa-SC + Pd; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel — Stratified on multiple myeloma (MM) isotype (immunoglobulin G [IgG] versus non-IgG), body weight (<=65 kg, >65 to <=85 kg, and >85 kg), and number of prior lines (1 to 2 versus >=3) according to IRT; Odds Ratio (OR) = 2.036, 95% CI 2-sided [1.425 to 2.908] — Two-sided 95% CI estimated using the Wald method

7. Secondary Outcome: Duration of Response (DOR)
Description: DOR: Time from the date of first response to the date of first occurrence of progressive disease (PD) determined by IRC or death from any cause, whichever occurred first.DOR was determined only for participants who achieved a response (PR or better).If PD/death not observed, participant was censored at date of last valid disease assessment performed prior to initiating further anti-myeloma treatment or analysis cut-off date, whichever occurred first. As per IMWG criteria: PD: increase of >=25% from lowest confirmed value in any 1 of following: serum M-protein (absolute increase>=0.5 gram/deciliter[g/dL]),serum M-protein increase>=1g/dL if lowest M-component >=5g/dL, urine M-component (absolute increase >=200mg/24h), appearance of new lesion(s),>=50% increase from nadir in SPD of >1 lesion or >=50% increase in longest diameter of a previous lesion >1 centimeter (cm) in short axis. PR: as defined in OM1.
Time Frame: From first dose of study medication administration (Day 1) up to PCD (06-Nov-2024), approximately 28 months
Population: The ITT population included all randomized population. Only responders (participants who achieved a response of PR or better subsequently confirmed based on disease assessment by IRC) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 187
months | NA [NA to NA] — NA indicates that median, lower and upper limit of CI were not estimable due to insufficient number of participants with events at PCD. | NA [18.300 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of participants with events at PCD.

8. Secondary Outcome: Time to First Response (TT1R)
Description: TT1R was defined as the time from randomization to the date of first IRC determined response (PR or better) that was subsequently confirmed. PR as per IMWG criteria was defined as >=50% reduction of serum M-protein and reduction in 24h urine M-protein by >=90% or to <200mg/24h. In addition to above, if present at baseline, >=50% reduction in the size SPD of STPs was also required.
Time Frame: From first dose of study medication administration (Day 1) up to PCD (06-Nov-2024), approximately 28 months
Population: The ITT population included all randomized population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 268 | 263
months | 1.91 [1.216 to 1.971] | 2.04 [1.906 to 2.793]

9. Secondary Outcome: Time to Best Response (TTBR)
Description: TTBR was defined as the time from randomization to the date of first occurrence of IRC determined best overall response (PR or better) that was subsequently confirmed. PR as per IMWG criteria was defined as >=50% reduction of serum M-protein and reduction in 24h urine M-protein by >=90% or to <200mg/24h. In addition to above, if present at baseline,>=50% reduction in the size SPD of STPs was also required.
Time Frame: From first dose of study medication administration (Day 1) up to PCD (06-Nov-2024), approximately 28 months
Population: The ITT population included all randomized population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 268 | 263
months | 3.94 [3.548 to 4.862] | 4.60 [3.811 to 5.125]

10. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization to the date of first documentation of PD as determined by IRC or the date of death from any cause, whichever came first. Responses will be determined according to IMWG criteria. PFS will be censored at the date of the last valid disease assessment not showing PD performed prior to initiation of a further anti-myeloma treatment (if any) or the analysis cut-off date, whichever comes first.
Time Frame: From first dose of study medication administration (Day 1) up to a maximum of 57 months
Reporting Status: Not Posted, anticipated posting 2028-03

11. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization to death from any cause. Participants without death prior to the analysis cut-off date will be censored at the last date the participant was known to be alive or the cut-off date, whichever is first.
Time Frame: From first dose of study medication administration (Day 1) up to a maximum of 57 months
Reporting Status: Not Posted, anticipated posting 2028-03

12. Secondary Outcome: Progression Free Survival 2 (PFS2)
Description: PFS2 is defined as time from the date of randomization to the date of first documentation of PD (as assessed by Investigator) after initiation of further anti-myeloma treatment or death from any cause, whichever happens first. Same censoring rule applies as in the PFS endpoint.
Time Frame: From first dose of study medication administration (Day 1) up to a maximum of 57 months
Reporting Status: Not Posted, anticipated posting 2028-03

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. SAEs were any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was a medically important event. TEAEs were defined as AEs that developed, worsened or became serious during the TE period.
Time Frame: From first dose of study medication administration (Day 1) up to 30 days after the last dose of study medication, approximately 28 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 264 | 263
Participants
  TEAEs | 255 | 255
  TESAEs | 127 | 139

14. Secondary Outcome: Isa-SC + Pd: Number of Participants With Injection Site Reactions (ISRs)
Description: The ISRs are defined as AEs related to medication administration with onset typically within 24 hours from the start of the infusion and are graded using NCI-CTCAE v5.0 criteria: Grade 1: tenderness with or without associated symptoms (warmth, erythema, itching). Grade 2: pain; lipodystrophy; edema; phlebitis. Grade 3: ulceration or necrosis severe tissue damage operative intervention indicated. Grade 4: life-threatening consequences; urgent intervention indicated. ISRs were collected through the eCRF. Number of participants with at least 1 ISR is reported. ISRs were applicable only for the SC administration.
Time Frame: as for outcome 13
Population: The safety population included ITT participants who received at least 1 dose or a part of a dose of the study medication. As pre-specified in the protocol and statistical analysis plan (SAP), ISRs were evaluated only for Isa-SC + Pd arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Isa-SC + Pd
Number analyzed (Participants) | 263
Participants | 11

15. Secondary Outcome: Ctrough of Isatuximab
Description: Plasma samples were collected at specified timepoints for the assessment of Ctrough.
Time Frame: Pre-dose on Cycle 1 Days 8, 15 and 22, Cycles 2 to 5 Days 1 and 15, Cycles 6, 7, 8, 9, 12, 15, 18, 21, 24 and 27 Day 1
Population: The PK population included all participants with at least 1 available isatuximab concentration post-baseline (whatever the cycle and even if dosing was incomplete) with adequate documentation of dosing and sampling dates and times. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 209 | 210
mcg/mL
  Cycle 1 Day 8: number analyzed (Participants) | 204 | 210
  Cycle 1 Day 8 | 92 (47) | 129 (66)
  Cycle 1 Day 15: number analyzed (Participants) | 179 | 187
  Cycle 1 Day 15 | 171 (84) | 249 (115)
  Cycle 1 Day 22: number analyzed (Participants) | 160 | 163
  Cycle 1 Day 22 | 227 (99) | 321 (144)
  Cycle 2 Day 1: number analyzed (Participants) | 140 | 147
  Cycle 2 Day 1 | 293 (117) | 407 (211)
  Cycle 2 Day 15: number analyzed (Participants) | 209 | 202
  Cycle 2 Day 15 | 243 (130) | 363 (228)
  Cycle 3 Day 1: number analyzed (Participants) | 179 | 160
  Cycle 3 Day 1 | 268 (133) | 381 (192)
  Cycle 3 Day 15: number analyzed (Participants) | 188 | 206
  Cycle 3 Day 15 | 256 (138) | 392 (245)
  Cycle 4 Day 1: number analyzed (Participants) | 167 | 167
  Cycle 4 Day 1 | 277 (151) | 477 (424)
  Cycle 4 Day 15: number analyzed (Participants) | 182 | 185
  Cycle 4 Day 15 | 285 (139) | 452 (400)
  Cycle 5 Day 1: number analyzed (Participants) | 156 | 153
  Cycle 5 Day 1 | 366 (568) | 470 (264)
  Cycle 5 Day 15: number analyzed (Participants) | 190 | 180
  Cycle 5 Day 15 | 306 (168) | 463 (275)
  Cycle 6 Day 1: number analyzed (Participants) | 158 | 145
  Cycle 6 Day 1 | 330 (165) | 491 (256)
  Cycle 7 Day 1: number analyzed (Participants) | 128 | 123
  Cycle 7 Day 1 | 339 (189) | 523 (336)
  Cycle 8 Day 1: number analyzed (Participants) | 116 | 100
  Cycle 8 Day 1 | 348 (172) | 569 (336)
  Cycle 9 Day 1: number analyzed (Participants) | 101 | 96
  Cycle 9 Day 1 | 365 (193) | 598 (369)
  Cycle 12 Day 1: number analyzed (Participants) | 63 | 63
  Cycle 12 Day 1 | 380 (214) | 593 (404)
  Cycle 15 Day 1: number analyzed (Participants) | 45 | 39
  Cycle 15 Day 1 | 354 (158) | 651 (361)
  Cycle 18 Day 1: number analyzed (Participants) | 18 | 23
  Cycle 18 Day 1 | 367 (140) | 645 (343)
  Cycle 21 Day 1: number analyzed (Participants) | 10 | 9
  Cycle 21 Day 1 | 388 (174) | 668 (213)
  Cycle 24 Day 1: number analyzed (Participants) | 2 | 3
  Cycle 24 Day 1 | 525 (455) | 651 (424)
  Cycle 27 Day 1: number analyzed (Participants) | 0 | 2
  Cycle 27 Day 1 |  | 566 (200)

16. Secondary Outcome: Isa-SC + Pd: Percentage of Successful Injections With Isatuximab Injector Device
Description: Percentage of successful injections with investigational isatuximab injector device was defined as completion of administration per provided instructions for use with no use errors or technical issues divided by the total number of injections x 100. Delivery performance of the device was analyzed based on the successful injection rate in the Isa-SC + Pd arm as the investigational isatuximab injector device was used only for SC administration.
Time Frame: From first dose of study medication administration (Day 1) up to PCD (06-Nov-2024), approximately 28 months
Population: The safety population included ITT participants who received at least 1 dose or a part of a dose of the study medication. Total number of actual injections is reported as type of units.
Measure: Number; unit: percentage of successful injections
Units Other Than Participants: Actual injections
Arm/Group | Isa-SC + Pd
Number analyzed (Participants) | 263
Number analyzed (Actual injections) | 5145
percentage of successful injections | 98.8

17. Secondary Outcome: Number of Participants With Treatment-emergent Anti-drug Antibodies (ADA) Against Isatuximab
Description: A participant with treatment-emergent ADA was a participant with at least 1 treatment induced or treatment boosted ADA at any time during the treatment or follow-up observation period. Treatment-induced ADA was defined as ADAs developed de novo (seroconversion) following administration of the biotherapeutic (ie, formation of ADAs any time after the initial study medication administration in a participant without pre-existing ADAs). Treatment-boosted ADA was defined as pre-existing ADAs that were boosted to a higher level following administration of biotherapeutic (ie, any time after the initial study medication administration) the ADA titer was significantly higher than the baseline titer. Number of participants with treatment-emergent ADAs is presented.
Time Frame: From first dose of study medication administration (Day 1) up to PCD (06-Nov-2024), approximately 28 months
Population: The ADA population included all participants from safety population with at least 1 ADA result (negative, positive or inconclusive) post-baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 254 | 255
Participants | 23 | 11

18. Secondary Outcome: Percentage of Participants With Response to 'Patient Expectation Questionnaire at Baseline (PEQ-BL)'
Description: Percentage of participants who responded that they strongly agree or agree at baseline with expectations of pain, discomfort and side effects from the injection method, the injection method would save time, study medication may result in side effects and would be worth taking are reported. PEQ-BL consisted of 7 items. Percentage of participants who ever received medication through IV and/or SC administration are also reported. Percentages are rounded off to the tenth decimal place. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: Baseline (Cycle 1 Day 1)
Population: The ITT population included all randomized population. Only those participants with data collected at Baseline are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 216 | 226
percentage of participants
  Injection method may be painful: strongly agree | 6.0 | 8.0
  Injection method may be painful: agree | 33.3 | 33.2
  Injection method may be uncomfortable: strongly agree | 11.1 | 9.7
  Injection method may be uncomfortable: agree | 37.5 | 26.1
  Injection method may result in side effects: strongly agree | 9.3 | 4.9
  Injection method may result in side effects: agree | 42.6 | 45.1
  Injection method will save me time: strongly agree | 9.3 | 21.2
  Injection method will save me time: agree | 31.5 | 51.8
  Study medication may result in side effects: strongly agree | 13.0 | 8.0
  Study medication may result in side effects: agree | 47.2 | 44.2
  Study medication would be worth taking: strongly agree | 26.9 | 27.0
  Study medication would be worth taking: agree | 46.8 | 47.8
  Ever received medication through IV | 74.1 | 61.9
  Ever received medication through SC | 48.6 | 61.1
  Neither received medication ever via IV or SC | 9.3 | 6.2

19. Secondary Outcome: Percentage of Participants Who Disagreed and Strongly Disagreed to 'PESQ-FU: Discomfort With Injection Method'
Description: The PESQ-FU consisting of 9 items has been designed to follow up on participant experience and satisfaction regarding the injection method (discomfort, pain, side effects, time saving and satisfaction) and study medication (side effects, worth taking, satisfaction and recommendation). This questionnaire has been adapted based on qualitative interviews with oncology participants. The responses to 'discomfort with injection method' were recorded as 'strongly agree, agree, neither agree nor disagree, disagree and strongly disagree' at specified timepoints. Percentage of participants who disagreed and strongly disagreed that they experienced any discomfort with the injection method are reported here. Percentages are rounded off to the tenth decimal place.
Time Frame: Cycle 1 Days 8, 15, 22, Cycle 2 Days 1 and 15, Cycles 3 and 4 Day 1, Cycles 5 to 29 Day 15
Population: The ITT population included all randomized population. Only those participants with data collected at specified timepoints are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 233 | 225
percentage of participants
  Cycle 1 Day 8: disagree: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: disagree | 33.5 | 39.5
  Cycle 1 Day 8: strongly disagree: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: strongly disagree | 14.7 | 36.8
  Cycle 1 Day 15: disagree: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: disagree | 38.9 | 43.3
  Cycle 1 Day 15: strongly disagree: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: strongly disagree | 14.9 | 37.9
  Cycle 1 Day 22: disagree: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: disagree | 39.8 | 44.2
  Cycle 1 Day 22: strongly disagree: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: strongly disagree | 12.8 | 33.0
  Cycle 2 Day 1: disagree | 40.8 | 48.9
  Cycle 2 Day 1: strongly disagree | 13.7 | 32.0
  Cycle 2 Day 15: disagree: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: disagree | 40.9 | 47.4
  Cycle 2 Day 15: strongly disagree: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: strongly disagree | 14.5 | 34.0
  Cycle 3 Day 1: disagree: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: disagree | 38.2 | 44.4
  Cycle 3 Day 1: strongly disagree: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: strongly disagree | 13.8 | 34.1
  Cycle 4 Day 1: disagree: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: disagree | 35.7 | 44.1
  Cycle 4 Day 1: strongly disagree: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: strongly disagree | 16.7 | 37.6
  Cycle 5 Day 15: disagree: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: disagree | 38.1 | 46.6
  Cycle 5 Day 15: strongly disagree: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: strongly disagree | 15.8 | 31.7
  Cycle 6 Day 15: disagree: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: disagree | 36.6 | 43.5
  Cycle 6 Day 15: strongly disagree: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: strongly disagree | 13.4 | 39.9
  Cycle 7 Day 15: disagree: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: disagree | 34.2 | 41.2
  Cycle 7 Day 15: strongly disagree: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: strongly disagree | 16.1 | 41.9
  Cycle 8 Day 15: disagree: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: disagree | 35.1 | 43.0
  Cycle 8 Day 15: strongly disagree: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: strongly disagree | 17.2 | 38.3
  Cycle 9 Day 15: disagree: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: disagree | 33.6 | 41.9
  Cycle 9 Day 15: strongly disagree: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: strongly disagree | 19.0 | 39.0
  Cycle 10 Day 15: disagree: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: disagree | 38.5 | 43.4
  Cycle 10 Day 15: strongly disagree: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: strongly disagree | 13.5 | 45.5
  Cycle 11 Day 15: disagree: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: disagree | 32.3 | 41.5
  Cycle 11 Day 15: strongly disagree: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: strongly disagree | 16.1 | 45.1
  Cycle 12 Day 15: disagree: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: disagree | 32.9 | 43.9
  Cycle 12 Day 15: strongly disagree: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: strongly disagree | 17.8 | 39.4
  Cycle 13 Day 15: disagree: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: disagree | 35.4 | 47.5
  Cycle 13 Day 15: strongly disagree: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: strongly disagree | 13.8 | 40.7
  Cycle 14 Day 15: disagree: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: disagree | 26.3 | 40.4
  Cycle 14 Day 15: strongly disagree: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: strongly disagree | 17.5 | 44.2
  Cycle 15 Day 15: disagree: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: disagree | 33.3 | 37.5
  Cycle 15 Day 15: strongly disagree: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: strongly disagree | 12.5 | 45.8
  Cycle 16 Day 15: disagree: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: disagree | 26.2 | 37.8
  Cycle 16 Day 15: strongly disagree: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: strongly disagree | 21.4 | 51.4
  Cycle 17 Day 15: disagree: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: disagree | 27.3 | 41.9
  Cycle 17 Day 15: strongly disagree: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: strongly disagree | 15.2 | 48.4
  Cycle 18 Day 15: disagree: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: disagree | 26.1 | 48.0
  Cycle 18 Day 15: strongly disagree: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: strongly disagree | 21.7 | 48.0
  Cycle 19 Day 15: disagree: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: disagree | 41.7 | 45.5
  Cycle 19 Day 15: strongly disagree: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: strongly disagree | 25.0 | 50.0
  Cycle 20 Day 15: disagree: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: disagree | 37.5 | 57.9
  Cycle 20 Day 15: strongly disagree: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: strongly disagree | 18.8 | 36.8
  Cycle 21 Day 15: disagree: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: disagree | 41.7 | 60.0
  Cycle 21 Day 15: strongly disagree: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: strongly disagree | 8.3 | 40.0
  Cycle 22 Day 15: disagree: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: disagree | 33.3 | 66.7
  Cycle 22 Day 15: strongly disagree: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: strongly disagree | 22.2 | 33.3
  Cycle 23 Day 15: disagree: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: disagree | 25.0 | 66.7
  Cycle 23 Day 15: strongly disagree: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: strongly disagree | 25.0 | 33.3
  Cycle 24 Day 15: disagree: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: disagree | 60.0 | 50.0
  Cycle 24 Day 15: strongly disagree: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: strongly disagree | 0 | 25.0
  Cycle 25 Day 15: disagree: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: disagree | 66.7 | 75.0
  Cycle 25 Day 15: strongly disagree: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: strongly disagree | 0 | 25.0
  Cycle 26 Day 15: disagree: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: disagree | 100 | 75.0
  Cycle 26 Day 15: strongly disagree: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: strongly disagree | 0 | 25.0
  Cycle 27 Day 15: disagree: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: disagree | 0 | 100
  Cycle 27 Day 15: strongly disagree: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: strongly disagree | 100 | 0
  Cycle 28 Day 15: disagree: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: disagree |  | 100
  Cycle 28 Day 15: strongly disagree: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: strongly disagree |  | 0
  Cycle 29 Day 15: disagree: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: disagree |  | 100
  Cycle 29 Day 15: strongly disagree: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: strongly disagree |  | 0

20. Secondary Outcome: Percentage of Participants Who Disagreed and Strongly Disagreed to 'PESQ-FU: Pain With Injection Method'
Description: The PESQ-FU consisting of 9 items has been designed to follow up on participant experience and satisfaction regarding the injection method (discomfort, pain, side effects, time saving and satisfaction) and study medication (side effects, worth taking, satisfaction and recommendation). This questionnaire has been adapted based on qualitative interviews with oncology participants. The responses to 'pain with injection method' were recorded as 'strongly agree, agree, neither agree nor disagree, disagree and strongly disagree' at specified timepoints. Percentage of participants who disagreed and strongly disagreed that they experienced any pain with the injection method are reported here. Percentages are rounded off to the tenth decimal place.
Time Frame: Cycle 1 Days 8, 15, 22, Cycle 2 Days 1 and 15, Cycles 3 and 4 Day 1, Cycles 5 to 29 Day 15
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 233 | 225
percentage of participants
  Cycle 1 Day 8: disagree: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: disagree | 44.5 | 42.7
  Cycle 1 Day 8: strongly disagree: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: strongly disagree | 20.2 | 40.9
  Cycle 1 Day 15: disagree: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: disagree | 47.6 | 44.3
  Cycle 1 Day 15: strongly disagree: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: strongly disagree | 18.8 | 40.4
  Cycle 1 Day 22: disagree: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: disagree | 43.6 | 45.6
  Cycle 1 Day 22: strongly disagree: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: strongly disagree | 19.4 | 36.9
  Cycle 2 Day 1: disagree | 48.9 | 51.6
  Cycle 2 Day 1: strongly disagree | 17.6 | 35.6
  Cycle 2 Day 15: disagree: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: disagree | 47.3 | 50.2
  Cycle 2 Day 15: strongly disagree: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: strongly disagree | 17.3 | 37.3
  Cycle 3 Day 1: disagree: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: disagree | 44.7 | 50.9
  Cycle 3 Day 1: strongly disagree: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: strongly disagree | 17.1 | 36.9
  Cycle 4 Day 1: disagree: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: disagree | 42.9 | 46.5
  Cycle 4 Day 1: strongly disagree: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: strongly disagree | 18.6 | 39.4
  Cycle 5 Day 15: disagree: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: disagree | 45.5 | 51.3
  Cycle 5 Day 15: strongly disagree: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: strongly disagree | 17.8 | 37.6
  Cycle 6 Day 15: disagree: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: disagree | 44.8 | 47.6
  Cycle 6 Day 15: strongly disagree: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: strongly disagree | 17.4 | 42.9
  Cycle 7 Day 15: disagree: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: disagree | 45.8 | 45.3
  Cycle 7 Day 15: strongly disagree: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: strongly disagree | 19.4 | 43.9
  Cycle 8 Day 15: disagree: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: disagree | 40.3 | 42.2
  Cycle 8 Day 15: strongly disagree: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: strongly disagree | 20.9 | 42.2
  Cycle 9 Day 15: disagree: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: disagree | 44.8 | 40.0
  Cycle 9 Day 15: strongly disagree: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: strongly disagree | 23.3 | 46.7
  Cycle 10 Day 15: disagree: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: disagree | 47.9 | 41.4
  Cycle 10 Day 15: strongly disagree: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: strongly disagree | 20.8 | 52.5
  Cycle 11 Day 15: disagree: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: disagree | 44.1 | 40.2
  Cycle 11 Day 15: strongly disagree: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: strongly disagree | 18.3 | 53.7
  Cycle 12 Day 15: disagree: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: disagree | 47.9 | 42.4
  Cycle 12 Day 15: strongly disagree: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: strongly disagree | 19.2 | 43.9
  Cycle 13 Day 15: disagree: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: disagree | 46.2 | 45.8
  Cycle 13 Day 15: strongly disagree: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: strongly disagree | 16.9 | 45.8
  Cycle 14 Day 15: disagree: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: disagree | 35.1 | 44.2
  Cycle 14 Day 15: strongly disagree: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: strongly disagree | 21.1 | 44.2
  Cycle 15 Day 15: disagree: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: disagree | 41.7 | 41.7
  Cycle 15 Day 15: strongly disagree: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: strongly disagree | 14.6 | 47.9
  Cycle 16 Day 15: disagree: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: disagree | 28.6 | 40.5
  Cycle 16 Day 15: strongly disagree: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: strongly disagree | 21.4 | 51.4
  Cycle 17 Day 15: disagree: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: disagree | 42.4 | 51.6
  Cycle 17 Day 15: strongly disagree: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: strongly disagree | 18.2 | 45.2
  Cycle 18 Day 15: disagree: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: disagree | 47.8 | 40.0
  Cycle 18 Day 15: strongly disagree: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: strongly disagree | 21.7 | 56.0
  Cycle 19 Day 15: disagree: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: disagree | 41.7 | 50.0
  Cycle 19 Day 15: strongly disagree: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: strongly disagree | 20.8 | 45.5
  Cycle 20 Day 15: disagree: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: disagree | 31.3 | 52.6
  Cycle 20 Day 15: strongly disagree: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: strongly disagree | 18.8 | 47.4
  Cycle 21 Day 15: disagree: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: disagree | 58.3 | 60.0
  Cycle 21 Day 15: strongly disagree: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: strongly disagree | 8.3 | 40.0
  Cycle 22 Day 15: disagree: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: disagree | 33.3 | 66.7
  Cycle 22 Day 15: strongly disagree: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: strongly disagree | 22.2 | 33.3
  Cycle 23 Day 15: disagree: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: disagree | 50.0 | 66.7
  Cycle 23 Day 15: strongly disagree: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: strongly disagree | 0 | 33.3
  Cycle 24 Day 15: disagree: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: disagree | 80.0 | 25.0
  Cycle 24 Day 15: strongly disagree: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: strongly disagree | 0 | 25.0
  Cycle 25 Day 15: disagree: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: disagree | 100 | 75.0
  Cycle 25 Day 15: strongly disagree: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: strongly disagree | 0 | 25.0
  Cycle 26 Day 15: disagree: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: disagree | 100 | 75.0
  Cycle 26 Day 15: strongly disagree: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: strongly disagree | 0 | 25.0
  Cycle 27 Day 15: disagree: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: disagree | 0 | 66.7
  Cycle 27 Day 15: strongly disagree: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: strongly disagree | 100 | 0
  Cycle 28 Day 15: disagree: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: disagree |  | 100
  Cycle 28 Day 15: strongly disagree: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: strongly disagree |  | 0
  Cycle 29 Day 15: disagree: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: disagree |  | 100
  Cycle 29 Day 15: strongly disagree: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: strongly disagree |  | 0

21. Secondary Outcome: Percentage of Participants Who Disagreed and Strongly Disagreed to 'PESQ-FU: Side Effects With Injection Method'
Description: The PESQ-FU consisting of 9 items has been designed to follow up on participant experience and satisfaction regarding the injection method (discomfort, pain, side effects, time saving and satisfaction) and study medication (side effects, worth taking, satisfaction and recommendation). This questionnaire has been adapted based on qualitative interviews with oncology participants. The responses to 'side effects with injection method' were recorded as 'strongly agree, agree, neither agree nor disagree, disagree and strongly disagree' at specified timepoints. Percentage of participants who disagreed and strongly disagreed that they experienced any side effects with the injection method are reported here. Percentages are rounded off to the tenth decimal place.
Time Frame: Cycle 1 Days 8, 15, 22, Cycle 2 Days 1 and 15, Cycles 3 and 4 Day 1, Cycles 5 to 29 Day 15
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 233 | 225
percentage of participants
  Cycle 1 Day 8: disagree: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: disagree | 41.3 | 46.8
  Cycle 1 Day 8: strongly disagree: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: strongly disagree | 17.9 | 28.2
  Cycle 1 Day 15: disagree: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: disagree | 40.4 | 46.3
  Cycle 1 Day 15: strongly disagree: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: strongly disagree | 15.4 | 25.1
  Cycle 1 Day 22: disagree: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: disagree | 44.5 | 42.7
  Cycle 1 Day 22: strongly disagree: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: strongly disagree | 12.3 | 23.3
  Cycle 2 Day 1: disagree | 45.9 | 51.1
  Cycle 2 Day 1: strongly disagree | 12.4 | 24.0
  Cycle 2 Day 15: disagree: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: disagree | 44.5 | 49.8
  Cycle 2 Day 15: strongly disagree: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: strongly disagree | 12.3 | 25.4
  Cycle 3 Day 1: disagree: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: disagree | 42.9 | 48.1
  Cycle 3 Day 1: strongly disagree: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: strongly disagree | 13.4 | 28.5
  Cycle 4 Day 1: disagree: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: disagree | 42.4 | 53.5
  Cycle 4 Day 1: strongly disagree: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: strongly disagree | 11.9 | 25.8
  Cycle 5 Day 15: disagree: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: disagree | 43.6 | 49.2
  Cycle 5 Day 15: strongly disagree: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: strongly disagree | 15.3 | 28.0
  Cycle 6 Day 15: disagree: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: disagree | 45.9 | 47.0
  Cycle 6 Day 15: strongly disagree: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: strongly disagree | 12.8 | 33.3
  Cycle 7 Day 15: disagree: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: disagree | 43.9 | 48.0
  Cycle 7 Day 15: strongly disagree: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: strongly disagree | 14.8 | 35.1
  Cycle 8 Day 15: disagree: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: disagree | 35.1 | 43.0
  Cycle 8 Day 15: strongly disagree: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: strongly disagree | 21.6 | 32.8
  Cycle 9 Day 15: disagree: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: disagree | 33.6 | 43.8
  Cycle 9 Day 15: strongly disagree: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: strongly disagree | 19.8 | 39.0
  Cycle 10 Day 15: disagree: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: disagree | 45.8 | 36.4
  Cycle 10 Day 15: strongly disagree: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: strongly disagree | 16.7 | 45.5
  Cycle 11 Day 15: disagree: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: disagree | 41.9 | 35.4
  Cycle 11 Day 15: strongly disagree: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: strongly disagree | 16.1 | 41.5
  Cycle 12 Day 15: disagree: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: disagree | 45.2 | 43.9
  Cycle 12 Day 15: strongly disagree: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: strongly disagree | 15.1 | 34.8
  Cycle 13 Day 15: disagree: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: disagree | 43.1 | 47.5
  Cycle 13 Day 15: strongly disagree: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: strongly disagree | 13.8 | 32.2
  Cycle 14 Day 15: disagree: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: disagree | 31.6 | 51.9
  Cycle 14 Day 15: strongly disagree: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: strongly disagree | 19.3 | 32.7
  Cycle 15 Day 15: disagree: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: disagree | 41.7 | 43.8
  Cycle 15 Day 15: strongly disagree: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: strongly disagree | 18.8 | 41.7
  Cycle 16 Day 15: disagree: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: disagree | 33.3 | 35.1
  Cycle 16 Day 15: strongly disagree: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: strongly disagree | 23.8 | 37.8
  Cycle 17 Day 15: disagree: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: disagree | 42.4 | 45.2
  Cycle 17 Day 15: strongly disagree: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: strongly disagree | 18.2 | 41.9
  Cycle 18 Day 15: disagree: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: disagree | 34.8 | 48.0
  Cycle 18 Day 15: strongly disagree: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: strongly disagree | 21.7 | 32.0
  Cycle 19 Day 15: disagree: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: disagree | 41.7 | 54.5
  Cycle 19 Day 15: strongly disagree: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: strongly disagree | 25.0 | 36.4
  Cycle 20 Day 15: disagree: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: disagree | 37.5 | 52.6
  Cycle 20 Day 15: strongly disagree: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: strongly disagree | 31.3 | 36.8
  Cycle 21 Day 15: disagree: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: disagree | 33.3 | 50.0
  Cycle 21 Day 15: strongly disagree: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: strongly disagree | 16.7 | 40.0
  Cycle 22 Day 15: disagree: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: disagree | 44.4 | 66.7
  Cycle 22 Day 15: strongly disagree: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: strongly disagree | 22.2 | 22.2
  Cycle 23 Day 15: disagree: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: disagree | 50.0 | 55.6
  Cycle 23 Day 15: strongly disagree: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: strongly disagree | 25.0 | 33.3
  Cycle 24 Day 15: disagree: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: disagree | 60.0 | 25.0
  Cycle 24 Day 15: strongly disagree: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: strongly disagree | 0 | 25.0
  Cycle 25 Day 15: disagree: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: disagree | 66.7 | 50.0
  Cycle 25 Day 15: strongly disagree: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: strongly disagree | 0 | 25.0
  Cycle 26 Day 15: disagree: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: disagree | 100 | 25.0
  Cycle 26 Day 15: strongly disagree: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: strongly disagree | 0 | 25.0
  Cycle 27 Day 15: disagree: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: disagree | 0 | 33.3
  Cycle 27 Day 15: strongly disagree: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: strongly disagree | 100 | 0
  Cycle 28 Day 15: disagree: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: disagree |  | 100
  Cycle 28 Day 15: strongly disagree: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: strongly disagree |  | 0
  Cycle 29 Day 15: disagree: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: disagree |  | 0
  Cycle 29 Day 15: strongly disagree: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: strongly disagree |  | 0

22. Secondary Outcome: Percentage of Participants Who Strongly Agreed and Agreed to 'PESQ-FU: Time Saving With Injection Method'
Description: The PESQ-FU consisting of 9 items has been designed to follow up on participant experience and satisfaction regarding the injection method (discomfort, pain, side effects, time saving and satisfaction) and study medication (side effects, worth taking, satisfaction and recommendation). This questionnaire has been adapted based on qualitative interviews with oncology participants. The responses to 'time saving with injection method' were recorded as 'strongly agree, agree, neither agree nor disagree, disagree and strongly disagree' at specified timepoints. Percentage of participants who strongly agreed and agreed that they experienced time saving with the injection method are reported here. Percentages are rounded off to the tenth decimal place.
Time Frame: Cycle 1 Days 8, 15, 22, Cycle 2 Days 1 and 15, Cycles 3 and 4 Day 1, Cycles 5 to 29 Day 15
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 233 | 225
percentage of participants
  Cycle 1 Day 8: strongly agree: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: strongly agree | 5.5 | 37.3
  Cycle 1 Day 8: agree: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: agree | 21.1 | 37.3
  Cycle 1 Day 15: strongly agree: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: strongly agree | 3.4 | 42.4
  Cycle 1 Day 15: agree: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: agree | 25.5 | 38.4
  Cycle 1 Day 22: strongly agree: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: strongly agree | 5.2 | 35.9
  Cycle 1 Day 22: agree: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: agree | 22.3 | 46.1
  Cycle 2 Day 1: strongly agree | 5.6 | 35.1
  Cycle 2 Day 1: agree | 25.8 | 46.2
  Cycle 2 Day 15: strongly agree: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: strongly agree | 5.5 | 33.0
  Cycle 2 Day 15: agree: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: agree | 28.2 | 48.3
  Cycle 3 Day 1: strongly agree: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: strongly agree | 3.7 | 39.3
  Cycle 3 Day 1: agree: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: agree | 25.8 | 46.3
  Cycle 4 Day 1: strongly agree: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: strongly agree | 7.6 | 37.6
  Cycle 4 Day 1: agree: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: agree | 22.4 | 43.7
  Cycle 5 Day 15: strongly agree: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: strongly agree | 9.9 | 39.7
  Cycle 5 Day 15: agree: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: agree | 22.8 | 43.4
  Cycle 6 Day 15: strongly agree: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: strongly agree | 7.6 | 39.9
  Cycle 6 Day 15: agree: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: agree | 28.5 | 39.9
  Cycle 7 Day 15: strongly agree: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: strongly agree | 7.7 | 41.9
  Cycle 7 Day 15: agree: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: agree | 29.0 | 40.5
  Cycle 8 Day 15: strongly agree: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: strongly agree | 12.7 | 35.2
  Cycle 8 Day 15: agree: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: agree | 23.9 | 45.3
  Cycle 9 Day 15: strongly agree: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: strongly agree | 10.3 | 47.6
  Cycle 9 Day 15: agree: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: agree | 26.7 | 34.3
  Cycle 10 Day 15: strongly agree: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: strongly agree | 9.4 | 42.4
  Cycle 10 Day 15: agree: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: agree | 26.0 | 35.4
  Cycle 11 Day 15: strongly agree: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: strongly agree | 6.5 | 45.1
  Cycle 11 Day 15: agree: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: agree | 33.3 | 37.8
  Cycle 12 Day 15: strongly agree: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: strongly agree | 11.0 | 36.4
  Cycle 12 Day 15: agree: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: agree | 26.0 | 42.4
  Cycle 13 Day 15: strongly agree: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: strongly agree | 9.2 | 44.1
  Cycle 13 Day 15: agree: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: agree | 26.2 | 42.4
  Cycle 14 Day 15: strongly agree: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: strongly agree | 12.3 | 42.3
  Cycle 14 Day 15: agree: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: agree | 14.0 | 40.4
  Cycle 15 Day 15: strongly agree: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: strongly agree | 14.6 | 41.7
  Cycle 15 Day 15: agree: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: agree | 16.7 | 50.0
  Cycle 16 Day 15: strongly agree: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: strongly agree | 16.7 | 48.6
  Cycle 16 Day 15: agree: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: agree | 26.2 | 37.8
  Cycle 17 Day 15: strongly agree: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: strongly agree | 18.2 | 51.6
  Cycle 17 Day 15: agree: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: agree | 24.2 | 35.5
  Cycle 18 Day 15: strongly agree: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: strongly agree | 26.1 | 56.0
  Cycle 18 Day 15: agree: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: agree | 26.1 | 32.0
  Cycle 19 Day 15: strongly agree: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: strongly agree | 20.8 | 50.0
  Cycle 19 Day 15: agree: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: agree | 16.7 | 40.9
  Cycle 20 Day 15: strongly agree: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: strongly agree | 12.5 | 52.6
  Cycle 20 Day 15: agree: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: agree | 25.0 | 36.8
  Cycle 21 Day 15: strongly agree: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: strongly agree | 16.7 | 50.0
  Cycle 21 Day 15: agree: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: agree | 33.3 | 30.0
  Cycle 22 Day 15: strongly agree: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: strongly agree | 11.1 | 33.3
  Cycle 22 Day 15: agree: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: agree | 55.6 | 44.4
  Cycle 23 Day 15: strongly agree: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: strongly agree | 25.0 | 33.3
  Cycle 23 Day 15: agree: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: agree | 75.0 | 44.4
  Cycle 24 Day 15: strongly agree: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: strongly agree | 0 | 25.0
  Cycle 24 Day 15: agree: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: agree | 80.0 | 50.0
  Cycle 25 Day 15: strongly agree: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: strongly agree | 0 | 25.0
  Cycle 25 Day 15: agree: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: agree | 66.7 | 50.0
  Cycle 26 Day 15: strongly agree: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: strongly agree | 0 | 50.0
  Cycle 26 Day 15: agree: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: agree | 100 | 25.0
  Cycle 27 Day 15: strongly agree: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: strongly agree | 0 | 0
  Cycle 27 Day 15: agree: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: agree | 100 | 66.7
  Cycle 28 Day 15: strongly agree: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: strongly agree |  | 0
  Cycle 28 Day 15: agree: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: agree |  | 50.0
  Cycle 29 Day 15: strongly agree: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: strongly agree |  | 0
  Cycle 29 Day 15: agree: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: agree |  | 0

23. Secondary Outcome: Percentage of Participants Who Responded Very Satisfied and Satisfied to 'PESQ-FU: Satisfaction With Injection Method'
Description: The PESQ-FU consisting of 9 items has been designed to follow up on participant experience and satisfaction regarding the injection method (discomfort, pain, side effects, time saving and satisfaction) and study medication (side effects, worth taking, satisfaction and recommendation). This questionnaire has been adapted based on qualitative interviews with oncology participants. The responses to 'satisfaction with injection method' were recorded as 'very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied and very dissatisfied' at specified timepoints. Percentage of participants who were very satisfied and satisfied with the injection method are reported here. Percentages are rounded off to the tenth decimal place.
Time Frame: Cycle 1 Days 8, 15, 22, Cycle 2 Days 1 and 15, Cycles 3 and 4 Day 1, Cycles 6 to 29 Day 15
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 233 | 225
percentage of participants
  Cycle 1 Day 8: very satisfied: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: very satisfied | 13.3 | 35.9
  Cycle 1 Day 8: satisfied: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: satisfied | 52.8 | 52.7
  Cycle 1 Day 15: very satisfied: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: very satisfied | 16.3 | 43.8
  Cycle 1 Day 15: satisfied: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: satisfied | 51.4 | 46.3
  Cycle 1 Day 22: very satisfied: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: very satisfied | 9.5 | 36.9
  Cycle 1 Day 22: satisfied: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: satisfied | 55.0 | 51.9
  Cycle 2 Day 1: very satisfied | 12.4 | 39.6
  Cycle 2 Day 1: satisfied | 51.9 | 48.4
  Cycle 2 Day 15: very satisfied: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: very satisfied | 14.5 | 40.2
  Cycle 2 Day 15: satisfied: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: satisfied | 54.5 | 51.7
  Cycle 3 Day 1: very satisfied: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: very satisfied | 13.4 | 42.1
  Cycle 3 Day 1: satisfied: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: satisfied | 57.6 | 48.1
  Cycle 4 Day 1: very satisfied: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: very satisfied | 13.8 | 43.2
  Cycle 4 Day 1: satisfied: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: satisfied | 55.7 | 50.7
  Cycle 6 Day 15: very satisfied: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: very satisfied | 14.5 | 45.8
  Cycle 6 Day 15: satisfied: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: satisfied | 54.1 | 47.0
  Cycle 7 Day 15: very satisfied: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: very satisfied | 17.4 | 50.0
  Cycle 7 Day 15: satisfied: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: satisfied | 54.8 | 45.3
  Cycle 8 Day 15: very satisfied: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: very satisfied | 18.7 | 45.3
  Cycle 8 Day 15: satisfied: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: satisfied | 49.3 | 45.3
  Cycle 9 Day 15: very satisfied: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: very satisfied | 20.7 | 51.4
  Cycle 9 Day 15: satisfied: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: satisfied | 50.0 | 43.8
  Cycle 10 Day 15: very satisfied: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: very satisfied | 16.7 | 52.5
  Cycle 10 Day 15: satisfied: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: satisfied | 49.0 | 41.4
  Cycle 11 Day 15: very satisfied: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: very satisfied | 19.4 | 56.1
  Cycle 11 Day 15: satisfied: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: satisfied | 48.4 | 40.2
  Cycle 12 Day 15: very satisfied: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: very satisfied | 17.8 | 48.5
  Cycle 12 Day 15: satisfied: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: satisfied | 49.3 | 45.5
  Cycle 13 Day 15: very satisfied: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: very satisfied | 23.1 | 50.8
  Cycle 13 Day 15: satisfied: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: satisfied | 50.8 | 45.8
  Cycle 14 Day 15: very satisfied: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: very satisfied | 24.6 | 50.0
  Cycle 14 Day 15: satisfied: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: satisfied | 43.9 | 42.3
  Cycle 15 Day 15: very satisfied: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: very satisfied | 27.1 | 56.3
  Cycle 15 Day 15: satisfied: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: satisfied | 37.5 | 39.6
  Cycle 16 Day 15: very satisfied: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: very satisfied | 28.6 | 54.1
  Cycle 16 Day 15: satisfied: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: satisfied | 45.2 | 45.9
  Cycle 17 Day 15: very satisfied: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: very satisfied | 27.3 | 51.6
  Cycle 17 Day 15: satisfied: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: satisfied | 45.5 | 41.9
  Cycle 18 Day 15: very satisfied: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: very satisfied | 26.1 | 60.0
  Cycle 18 Day 15: satisfied: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: satisfied | 52.2 | 36.0
  Cycle 19 Day 15: very satisfied: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: very satisfied | 29.2 | 50.0
  Cycle 19 Day 15: satisfied: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: satisfied | 45.8 | 50.0
  Cycle 20 Day 15: very satisfied: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: very satisfied | 31.3 | 52.6
  Cycle 20 Day 15: satisfied: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: satisfied | 43.8 | 42.1
  Cycle 21 Day 15: very satisfied: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: very satisfied | 25.0 | 80.0
  Cycle 21 Day 15: satisfied: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: satisfied | 41.7 | 20.0
  Cycle 22 Day 15: very satisfied: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: very satisfied | 55.6 | 44.4
  Cycle 22 Day 15: satisfied: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: satisfied | 33.3 | 55.6
  Cycle 23 Day 15: very satisfied: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: very satisfied | 50.0 | 55.6
  Cycle 23 Day 15: satisfied: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: satisfied | 50.0 | 44.4
  Cycle 24 Day 15: very satisfied: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: very satisfied | 40.0 | 50.0
  Cycle 24 Day 15: satisfied: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: satisfied | 40.0 | 50.0
  Cycle 25 Day 15: very satisfied: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: very satisfied | 0 | 50.0
  Cycle 25 Day 15: satisfied: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: satisfied | 100 | 50.0
  Cycle 26 Day 15: very satisfied: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: very satisfied | 50.0 | 75.0
  Cycle 26 Day 15: satisfied: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: satisfied | 50.0 | 25.0
  Cycle 27 Day 15: very satisfied: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: very satisfied | 0 | 33.3
  Cycle 27 Day 15: satisfied: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: satisfied | 100 | 66.7
  Cycle 28 Day 15: very satisfied: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: very satisfied |  | 50.0
  Cycle 28 Day 15: satisfied: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: satisfied |  | 50.0
  Cycle 29 Day 15: very satisfied: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: very satisfied |  | 0
  Cycle 29 Day 15: satisfied: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: satisfied |  | 100

24. Secondary Outcome: Percentage of Participants Who Disagreed and Strongly Disagreed to 'PESQ-FU: Side Effects With Study Medication'
Description: The PESQ-FU consisting of 9 items has been designed to follow up on participant experience and satisfaction regarding the injection method (discomfort, pain, side effects, time saving and satisfaction) and study medication (side effects, worth taking, satisfaction and recommendation). This questionnaire has been adapted based on qualitative interviews with oncology participants. The responses to 'side effects with study medication' were recorded as 'strongly agree, agree, neither agree nor disagree, disagree and strongly disagree' at specified timepoints. Percentage of participants who disagreed and strongly disagreed that they experienced any side effects with study medication are reported here. Percentages are rounded off to the tenth decimal place.
Time Frame: Cycle 1 Days 8, 15, 22, Cycle 2 Days 1 and 15, Cycles 3 and 4 Day 1, Cycles 5 to 29 Day 15
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 233 | 225
percentage of participants
  Cycle 1 Day 8: disagree: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: disagree | 35.3 | 44.5
  Cycle 1 Day 8: strongly disagree: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: strongly disagree | 16.1 | 25.0
  Cycle 1 Day 15: disagree: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: disagree | 38.0 | 38.9
  Cycle 1 Day 15: strongly disagree: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: strongly disagree | 13.0 | 23.6
  Cycle 1 Day 22: disagree: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: disagree | 41.2 | 40.3
  Cycle 1 Day 22: strongly disagree: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: strongly disagree | 9.0 | 19.9
  Cycle 2 Day 1: disagree | 37.8 | 46.7
  Cycle 2 Day 1: strongly disagree | 9.4 | 23.1
  Cycle 2 Day 15: disagree: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: disagree | 41.4 | 47.8
  Cycle 2 Day 15: strongly disagree: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: strongly disagree | 10.5 | 20.1
  Cycle 3 Day 1: disagree: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: disagree | 40.6 | 40.7
  Cycle 3 Day 1: strongly disagree: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: strongly disagree | 11.1 | 27.1
  Cycle 4 Day 1: disagree: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: disagree | 39.0 | 48.8
  Cycle 4 Day 1: strongly disagree: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: strongly disagree | 11.4 | 23.0
  Cycle 5 Day 15: disagree: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: disagree | 39.1 | 46.6
  Cycle 5 Day 15: strongly disagree: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: strongly disagree | 12.9 | 25.9
  Cycle 6 Day 15: disagree: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: disagree | 39.5 | 44.6
  Cycle 6 Day 15: strongly disagree: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: strongly disagree | 13.4 | 28.6
  Cycle 7 Day 15: disagree: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: disagree | 39.4 | 41.2
  Cycle 7 Day 15: strongly disagree: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: strongly disagree | 14.8 | 34.5
  Cycle 8 Day 15: disagree: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: disagree | 33.6 | 38.3
  Cycle 8 Day 15: strongly disagree: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: strongly disagree | 17.2 | 31.3
  Cycle 9 Day 15: disagree: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: disagree | 31.0 | 43.8
  Cycle 9 Day 15: strongly disagree: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: strongly disagree | 17.2 | 33.3
  Cycle 10 Day 15: disagree: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: disagree | 39.6 | 36.4
  Cycle 10 Day 15: strongly disagree: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: strongly disagree | 15.6 | 41.4
  Cycle 11 Day 15: disagree: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: disagree | 38.7 | 31.7
  Cycle 11 Day 15: strongly disagree: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: strongly disagree | 16.1 | 39.0
  Cycle 12 Day 15: disagree: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: disagree | 37.0 | 42.4
  Cycle 12 Day 15: strongly disagree: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: strongly disagree | 15.1 | 31.8
  Cycle 13 Day 15: disagree: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: disagree | 40.0 | 39.0
  Cycle 13 Day 15: strongly disagree: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: strongly disagree | 15.4 | 33.9
  Cycle 14 Day 15: disagree: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: disagree | 33.3 | 50.0
  Cycle 14 Day 15: strongly disagree: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: strongly disagree | 19.3 | 28.8
  Cycle 15 Day 15: disagree: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: disagree | 35.4 | 39.6
  Cycle 15 Day 15: strongly disagree: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: strongly disagree | 22.9 | 41.7
  Cycle 16 Day 15: disagree: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: disagree | 31.0 | 29.7
  Cycle 16 Day 15: strongly disagree: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: strongly disagree | 23.8 | 40.5
  Cycle 17 Day 15: disagree: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: disagree | 27.3 | 45.2
  Cycle 17 Day 15: strongly disagree: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: strongly disagree | 27.3 | 35.5
  Cycle 18 Day 15: disagree: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: disagree | 26.1 | 48.0
  Cycle 18 Day 15: strongly disagree: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: strongly disagree | 34.8 | 36.0
  Cycle 19 Day 15: disagree: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: disagree | 25.0 | 50.0
  Cycle 19 Day 15: strongly disagree: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: strongly disagree | 25.0 | 31.8
  Cycle 20 Day 15: disagree: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: disagree | 18.8 | 57.9
  Cycle 20 Day 15: strongly disagree: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: strongly disagree | 31.3 | 26.3
  Cycle 21 Day 15: disagree: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: disagree | 25.0 | 60.0
  Cycle 21 Day 15: strongly disagree: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: strongly disagree | 16.7 | 30.0
  Cycle 22 Day 15: disagree: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: disagree | 44.4 | 55.6
  Cycle 22 Day 15: strongly disagree: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: strongly disagree | 22.2 | 33.3
  Cycle 23 Day 15: disagree: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: disagree | 50.0 | 44.4
  Cycle 23 Day 15: strongly disagree: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: strongly disagree | 25.0 | 33.3
  Cycle 24 Day 15: disagree: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: disagree | 40.0 | 25.0
  Cycle 24 Day 15: strongly disagree: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: strongly disagree | 0 | 25.0
  Cycle 25 Day 15: disagree: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: disagree | 66.7 | 50.0
  Cycle 25 Day 15: strongly disagree: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: strongly disagree | 0 | 25.0
  Cycle 26 Day 15: disagree: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: disagree | 100 | 25.0
  Cycle 26 Day 15: strongly disagree: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: strongly disagree | 0 | 25.0
  Cycle 27 Day 15: disagree: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: disagree | 0 | 33.3
  Cycle 27 Day 15: strongly disagree: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: strongly disagree | 100 | 0
  Cycle 28 Day 15: disagree: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: disagree |  | 50.0
  Cycle 28 Day 15: strongly disagree: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: strongly disagree |  | 0
  Cycle 29 Day 15: disagree: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: disagree |  | 0
  Cycle 29 Day 15: strongly disagree: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: strongly disagree |  | 0

25. Secondary Outcome: Percentage of Participants Who Strongly Agreed and Agreed to 'PESQ-FU: Study Medication Worth Taking'
Description: The PESQ-FU consisting of 9 items has been designed to follow up on participant experience and satisfaction regarding the injection method (discomfort, pain, side effects, time saving and satisfaction) and study medication (side effects, worth taking, satisfaction and recommendation). This questionnaire has been adapted based on qualitative interviews with oncology participants. The responses to 'study medication worth taking' were recorded as 'strongly agree, agree, neither agree nor disagree, disagree and strongly disagree' at specified timepoints. Percentage of participants who strongly agreed and agreed that the study medication was worth taking are reported here. Percentages are rounded off to the tenth decimal place.
Time Frame: Cycle 1 Days 8, 15, 22, Cycle 2 Days 1 and 15, Cycles 3 and 4 Day 1, Cycles 5 to 29 Day 15
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 233 | 225
percentage of participants
  Cycle 1 Day 8: strongly agree: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: strongly agree | 17.9 | 34.1
  Cycle 1 Day 8: agree: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: agree | 48.6 | 42.3
  Cycle 1 Day 15: strongly agree: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: strongly agree | 19.7 | 33.0
  Cycle 1 Day 15: agree: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: agree | 51.4 | 48.8
  Cycle 1 Day 22: strongly agree: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: strongly agree | 20.9 | 30.6
  Cycle 1 Day 22: agree: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: agree | 45.5 | 47.1
  Cycle 2 Day 1: strongly agree | 21.0 | 34.2
  Cycle 2 Day 1: agree | 48.9 | 47.1
  Cycle 2 Day 15: strongly agree: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: strongly agree | 21.4 | 32.1
  Cycle 2 Day 15: agree: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: agree | 50.5 | 50.7
  Cycle 3 Day 1: strongly agree: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: strongly agree | 20.7 | 43.0
  Cycle 3 Day 1: agree: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: agree | 53.0 | 46.3
  Cycle 4 Day 1: strongly agree: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: strongly agree | 22.9 | 39.0
  Cycle 4 Day 1: agree: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: agree | 54.8 | 47.4
  Cycle 5 Day 15: strongly agree: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: strongly agree | 25.2 | 42.9
  Cycle 5 Day 15: agree: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: agree | 49.5 | 50.3
  Cycle 6 Day 15: strongly agree: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: strongly agree | 25.0 | 41.1
  Cycle 6 Day 15: agree: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: agree | 50.6 | 48.8
  Cycle 7 Day 15: strongly agree: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: strongly agree | 25.2 | 45.3
  Cycle 7 Day 15: agree: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: agree | 56.1 | 44.6
  Cycle 8 Day 15: strongly agree: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: strongly agree | 26.9 | 40.6
  Cycle 8 Day 15: agree: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: agree | 52.2 | 50.0
  Cycle 9 Day 15: strongly agree: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: strongly agree | 30.2 | 43.8
  Cycle 9 Day 15: agree: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: agree | 49.1 | 46.7
  Cycle 10 Day 15: strongly agree: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: strongly agree | 25.0 | 45.5
  Cycle 10 Day 15: agree: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: agree | 51.0 | 46.5
  Cycle 11 Day 15: strongly agree: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: strongly agree | 24.7 | 52.4
  Cycle 11 Day 15: agree: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: agree | 54.8 | 36.6
  Cycle 12 Day 15: strongly agree: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: strongly agree | 28.8 | 43.9
  Cycle 12 Day 15: agree: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: agree | 56.2 | 47.0
  Cycle 13 Day 15: strongly agree: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: strongly agree | 32.3 | 40.7
  Cycle 13 Day 15: agree: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: agree | 49.2 | 54.2
  Cycle 14 Day 15: strongly agree: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: strongly agree | 40.4 | 42.3
  Cycle 14 Day 15: agree: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: agree | 36.8 | 50.0
  Cycle 15 Day 15: strongly agree: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: strongly agree | 35.4 | 54.2
  Cycle 15 Day 15: agree: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: agree | 41.7 | 39.6
  Cycle 16 Day 15: strongly agree: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: strongly agree | 42.9 | 45.9
  Cycle 16 Day 15: agree: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: agree | 38.1 | 48.6
  Cycle 17 Day 15: strongly agree: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: strongly agree | 51.5 | 51.6
  Cycle 17 Day 15: agree: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: agree | 30.3 | 45.2
  Cycle 18 Day 15: strongly agree: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: strongly agree | 47.8 | 60.0
  Cycle 18 Day 15: agree: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: agree | 34.8 | 40.0
  Cycle 19 Day 15: strongly agree: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: strongly agree | 45.8 | 54.5
  Cycle 19 Day 15: agree: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: agree | 33.3 | 40.9
  Cycle 20 Day 15: strongly agree: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: strongly agree | 43.8 | 63.2
  Cycle 20 Day 15: agree: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: agree | 25.0 | 36.8
  Cycle 21 Day 15: strongly agree: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: strongly agree | 50.0 | 50.0
  Cycle 21 Day 15: agree: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: agree | 25.0 | 50.0
  Cycle 22 Day 15: strongly agree: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: strongly agree | 66.7 | 33.3
  Cycle 22 Day 15: agree: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: agree | 22.2 | 66.7
  Cycle 23 Day 15: strongly agree: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: strongly agree | 75.0 | 55.6
  Cycle 23 Day 15: agree: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: agree | 25.0 | 44.4
  Cycle 24 Day 15: strongly agree: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: strongly agree | 40.0 | 50.0
  Cycle 24 Day 15: agree: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: agree | 60.0 | 50.0
  Cycle 25 Day 15: strongly agree: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: strongly agree | 33.3 | 50.0
  Cycle 25 Day 15: agree: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: agree | 66.7 | 50.0
  Cycle 26 Day 15: strongly agree: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: strongly agree | 50.0 | 75.0
  Cycle 26 Day 15: agree: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: agree | 50.0 | 25.0
  Cycle 27 Day 15: strongly agree: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: strongly agree | 0 | 33.3
  Cycle 27 Day 15: agree: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: agree | 100 | 66.7
  Cycle 28 Day 15: strongly agree: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: strongly agree |  | 50.0
  Cycle 28 Day 15: agree: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: agree |  | 50.0
  Cycle 29 Day 15: strongly agree: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: strongly agree |  | 0
  Cycle 29 Day 15: agree: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: agree |  | 100

26. Secondary Outcome: Percentage of Participants Who Responded Very Satisfied and Satisfied to 'PESQ-FU: Satisfaction With Study Medication'
Description: The PESQ-FU consisting of 9 items has been designed to follow up on participant experience and satisfaction regarding the injection method (discomfort, pain, side effects, time saving and satisfaction) and study medication (side effects, worth taking, satisfaction and recommendation). This questionnaire has been adapted based on qualitative interviews with oncology participants. The responses to satisfaction with study medication were recorded as 'very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied and very dissatisfied' at specified timepoints. Percentage of participants who were very satisfied and satisfied with the study medication are reported here. Percentages are rounded off to the tenth decimal place.
Time Frame: Cycle 1 Days 8, 15, 22, Cycle 2 Days 1 and 15, Cycles 3 and 4 Day 1, Cycles 5 to 29 Day 15
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 233 | 225
percentage of participants
  Cycle 1 Day 8: very satisfied: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: very satisfied | 17.0 | 29.5
  Cycle 1 Day 8: satisfied: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: satisfied | 56.0 | 50.5
  Cycle 1 Day 15: very satisfied: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: very satisfied | 21.2 | 31.0
  Cycle 1 Day 15: satisfied: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: satisfied | 47.6 | 47.8
  Cycle 1 Day 22: very satisfied: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: very satisfied | 15.6 | 30.6
  Cycle 1 Day 22: satisfied: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: satisfied | 58.3 | 48.1
  Cycle 2 Day 1: very satisfied | 18.9 | 31.1
  Cycle 2 Day 1: satisfied | 53.6 | 50.2
  Cycle 2 Day 15: very satisfied: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: very satisfied | 20.5 | 30.6
  Cycle 2 Day 15: satisfied: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: satisfied | 57.3 | 52.2
  Cycle 3 Day 1: very satisfied: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: very satisfied | 18.9 | 38.3
  Cycle 3 Day 1: satisfied: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: satisfied | 61.8 | 49.5
  Cycle 4 Day 1: very satisfied: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: very satisfied | 21.0 | 38.0
  Cycle 4 Day 1: satisfied: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: satisfied | 60.0 | 50.2
  Cycle 5 Day 15: very satisfied: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: very satisfied | 27.2 | 46.0
  Cycle 5 Day 15: satisfied: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: satisfied | 55.0 | 46.0
  Cycle 6 Day 15: very satisfied: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: very satisfied | 26.2 | 41.7
  Cycle 6 Day 15: satisfied: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: satisfied | 56.4 | 46.4
  Cycle 7 Day 15: very satisfied: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: very satisfied | 30.3 | 45.9
  Cycle 7 Day 15: satisfied: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: satisfied | 52.3 | 47.3
  Cycle 8 Day 15: very satisfied: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: very satisfied | 29.9 | 43.8
  Cycle 8 Day 15: satisfied: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: satisfied | 55.2 | 46.9
  Cycle 9 Day 15: very satisfied: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: very satisfied | 35.3 | 48.6
  Cycle 9 Day 15: satisfied: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: satisfied | 50.0 | 43.8
  Cycle 10 Day 15: very satisfied: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: very satisfied | 32.3 | 49.5
  Cycle 10 Day 15: satisfied: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: satisfied | 50.0 | 43.4
  Cycle 11 Day 15: very satisfied: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: very satisfied | 29.0 | 50.0
  Cycle 11 Day 15: satisfied: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: satisfied | 58.1 | 42.7
  Cycle 12 Day 15: very satisfied: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: very satisfied | 28.8 | 39.4
  Cycle 12 Day 15: satisfied: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: satisfied | 56.2 | 48.5
  Cycle 13 Day 15: very satisfied: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: very satisfied | 36.9 | 49.2
  Cycle 13 Day 15: satisfied: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: satisfied | 47.7 | 42.4
  Cycle 14 Day 15: very satisfied: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: very satisfied | 42.1 | 46.2
  Cycle 14 Day 15: satisfied: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: satisfied | 45.6 | 44.2
  Cycle 15 Day 15: very satisfied: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: very satisfied | 41.7 | 56.3
  Cycle 15 Day 15: satisfied: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: satisfied | 43.8 | 37.5
  Cycle 16 Day 15: very satisfied: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: very satisfied | 45.2 | 48.6
  Cycle 16 Day 15: satisfied: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: satisfied | 35.7 | 45.9
  Cycle 17 Day 15: very satisfied: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: very satisfied | 45.5 | 51.6
  Cycle 17 Day 15: satisfied: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: satisfied | 39.4 | 45.2
  Cycle 18 Day 15: very satisfied: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: very satisfied | 43.5 | 68.0
  Cycle 18 Day 15: satisfied: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: satisfied | 43.5 | 28.0
  Cycle 19 Day 15: very satisfied: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: very satisfied | 37.5 | 59.1
  Cycle 19 Day 15: satisfied: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: satisfied | 41.7 | 36.4
  Cycle 20 Day 15: very satisfied: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: very satisfied | 50.0 | 42.1
  Cycle 20 Day 15: satisfied: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: satisfied | 25.0 | 52.6
  Cycle 21 Day 15: very satisfied: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: very satisfied | 50.0 | 80.0
  Cycle 21 Day 15: satisfied: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: satisfied | 25.0 | 20.0
  Cycle 22 Day 15: very satisfied: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: very satisfied | 66.7 | 33.3
  Cycle 22 Day 15: satisfied: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: satisfied | 22.2 | 66.7
  Cycle 23 Day 15: very satisfied: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: very satisfied | 50.0 | 55.6
  Cycle 23 Day 15: satisfied: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: satisfied | 50.0 | 44.4
  Cycle 24 Day 15: very satisfied: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: very satisfied | 80.0 | 50.0
  Cycle 24 Day 15: satisfied: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: satisfied | 0 | 25.0
  Cycle 25 Day 15: very satisfied: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: very satisfied | 33.3 | 50.0
  Cycle 25 Day 15: satisfied: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: satisfied | 33.3 | 50.0
  Cycle 26 Day 15: very satisfied: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: very satisfied | 50.0 | 75.0
  Cycle 26 Day 15: satisfied: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: satisfied | 50.0 | 25.0
  Cycle 27 Day 15: very satisfied: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: very satisfied | 0 | 66.7
  Cycle 27 Day 15: satisfied: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: satisfied | 100 | 33.3
  Cycle 28 Day 15: very satisfied: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: very satisfied |  | 50.0
  Cycle 28 Day 15: satisfied: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: satisfied |  | 50.0
  Cycle 29 Day 15: very satisfied: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: very satisfied |  | 0
  Cycle 29 Day 15: satisfied: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: satisfied |  | 100

27. Secondary Outcome: Percentage of Participants Who Responded Definitely Yes and Probably Yes to 'PESQ-FU: Recommendation of Study Medication'
Description: The PESQ-FU consisting of 9 items has been designed to follow up on participant experience and satisfaction regarding the injection method (discomfort, pain, side effects, time saving and satisfaction) and study medication (side effects, worth taking, satisfaction and recommendation). This questionnaire has been adapted based on qualitative interviews with oncology participants. The responses to 'recommendation of the study medication' were recorded as 'definitely yes, probably yes, unsure, probably not and definitely not' at specified timepoints. Percentage of participants who responded definitely yes and probably yes to the recommendation of study medication are reported here. Percentages are rounded off to the tenth decimal place.
Time Frame: Cycle 1 Days 8, 15, 22, Cycle 2 Days 1 and 15, Cycles 3 and 4 Day 1, Cycles 5 to 29 Day 15
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 233 | 225
percentage of participants
  Cycle 1 Day 8: definitely yes: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: definitely yes | 24.8 | 50.9
  Cycle 1 Day 8: probably yes: number analyzed (Participants) | 218 | 220
  Cycle 1 Day 8: probably yes | 43.1 | 34.1
  Cycle 1 Day 15: definitely yes: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: definitely yes | 29.3 | 46.8
  Cycle 1 Day 15: probably yes: number analyzed (Participants) | 208 | 203
  Cycle 1 Day 15: probably yes | 44.7 | 36.9
  Cycle 1 Day 22: definitely yes: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: definitely yes | 26.5 | 46.6
  Cycle 1 Day 22: probably yes: number analyzed (Participants) | 211 | 206
  Cycle 1 Day 22: probably yes | 46.9 | 38.8
  Cycle 2 Day 1: definitely yes | 25.8 | 49.8
  Cycle 2 Day 1: probably yes | 42.9 | 36.4
  Cycle 2 Day 15: definitely yes: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: definitely yes | 26.8 | 46.9
  Cycle 2 Day 15: probably yes: number analyzed (Participants) | 220 | 209
  Cycle 2 Day 15: probably yes | 46.8 | 39.2
  Cycle 3 Day 1: definitely yes: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: definitely yes | 28.1 | 52.8
  Cycle 3 Day 1: probably yes: number analyzed (Participants) | 217 | 214
  Cycle 3 Day 1: probably yes | 48.8 | 37.4
  Cycle 4 Day 1: definitely yes: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: definitely yes | 29.5 | 53.1
  Cycle 4 Day 1: probably yes: number analyzed (Participants) | 210 | 213
  Cycle 4 Day 1: probably yes | 50.0 | 38.5
  Cycle 5 Day 15: definitely yes: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: definitely yes | 33.7 | 58.7
  Cycle 5 Day 15: probably yes: number analyzed (Participants) | 202 | 189
  Cycle 5 Day 15: probably yes | 48.0 | 34.9
  Cycle 6 Day 15: definitely yes: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: definitely yes | 33.7 | 57.1
  Cycle 6 Day 15: probably yes: number analyzed (Participants) | 172 | 168
  Cycle 6 Day 15: probably yes | 45.9 | 38.1
  Cycle 7 Day 15: definitely yes: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: definitely yes | 30.3 | 58.1
  Cycle 7 Day 15: probably yes: number analyzed (Participants) | 155 | 148
  Cycle 7 Day 15: probably yes | 47.7 | 36.5
  Cycle 8 Day 15: definitely yes: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: definitely yes | 39.6 | 55.5
  Cycle 8 Day 15: probably yes: number analyzed (Participants) | 134 | 128
  Cycle 8 Day 15: probably yes | 38.8 | 37.5
  Cycle 9 Day 15: definitely yes: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: definitely yes | 36.2 | 60.0
  Cycle 9 Day 15: probably yes: number analyzed (Participants) | 116 | 105
  Cycle 9 Day 15: probably yes | 43.1 | 37.1
  Cycle 10 Day 15: definitely yes: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: definitely yes | 37.5 | 60.6
  Cycle 10 Day 15: probably yes: number analyzed (Participants) | 96 | 99
  Cycle 10 Day 15: probably yes | 41.7 | 34.3
  Cycle 11 Day 15: definitely yes: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: definitely yes | 35.5 | 64.6
  Cycle 11 Day 15: probably yes: number analyzed (Participants) | 93 | 82
  Cycle 11 Day 15: probably yes | 38.7 | 29.3
  Cycle 12 Day 15: definitely yes: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: definitely yes | 31.5 | 51.5
  Cycle 12 Day 15: probably yes: number analyzed (Participants) | 73 | 66
  Cycle 12 Day 15: probably yes | 34.2 | 40.9
  Cycle 13 Day 15: definitely yes: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: definitely yes | 35.4 | 62.7
  Cycle 13 Day 15: probably yes: number analyzed (Participants) | 65 | 59
  Cycle 13 Day 15: probably yes | 35.4 | 32.2
  Cycle 14 Day 15: definitely yes: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: definitely yes | 33.3 | 61.5
  Cycle 14 Day 15: probably yes: number analyzed (Participants) | 57 | 52
  Cycle 14 Day 15: probably yes | 31.6 | 32.7
  Cycle 15 Day 15: definitely yes: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: definitely yes | 41.7 | 64.6
  Cycle 15 Day 15: probably yes: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15: probably yes | 31.3 | 27.1
  Cycle 16 Day 15: definitely yes: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: definitely yes | 42.9 | 56.8
  Cycle 16 Day 15: probably yes: number analyzed (Participants) | 42 | 37
  Cycle 16 Day 15: probably yes | 28.6 | 35.1
  Cycle 17 Day 15: definitely yes: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: definitely yes | 51.5 | 54.8
  Cycle 17 Day 15: probably yes: number analyzed (Participants) | 33 | 31
  Cycle 17 Day 15: probably yes | 12.1 | 38.7
  Cycle 18 Day 15: definitely yes: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: definitely yes | 43.5 | 68.0
  Cycle 18 Day 15: probably yes: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15: probably yes | 21.7 | 28.0
  Cycle 19 Day 15: definitely yes: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: definitely yes | 45.8 | 63.6
  Cycle 19 Day 15: probably yes: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15: probably yes | 25.0 | 36.4
  Cycle 20 Day 15: definitely yes: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: definitely yes | 56.3 | 68.4
  Cycle 20 Day 15: probably yes: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15: probably yes | 18.8 | 26.3
  Cycle 21 Day 15: definitely yes: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: definitely yes | 50.0 | 60.0
  Cycle 21 Day 15: probably yes: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15: probably yes | 25.0 | 30.0
  Cycle 22 Day 15: definitely yes: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: definitely yes | 66.7 | 44.4
  Cycle 22 Day 15: probably yes: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15: probably yes | 22.2 | 44.4
  Cycle 23 Day 15: definitely yes: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: definitely yes | 75.0 | 66.7
  Cycle 23 Day 15: probably yes: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15: probably yes | 25.0 | 22.2
  Cycle 24 Day 15: definitely yes: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: definitely yes | 60.0 | 50.0
  Cycle 24 Day 15: probably yes: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15: probably yes | 20.0 | 25.0
  Cycle 25 Day 15: definitely yes: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: definitely yes | 33.3 | 50.0
  Cycle 25 Day 15: probably yes: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15: probably yes | 66.7 | 25.0
  Cycle 26 Day 15: definitely yes: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: definitely yes | 50.0 | 50.0
  Cycle 26 Day 15: probably yes: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15: probably yes | 50.0 | 25.0
  Cycle 27 Day 15: definitely yes: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: definitely yes | 100 | 33.3
  Cycle 27 Day 15: probably yes: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15: probably yes | 0 | 33.3
  Cycle 28 Day 15: definitely yes: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: definitely yes |  | 50.0
  Cycle 28 Day 15: probably yes: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15: probably yes |  | 0
  Cycle 29 Day 15: definitely yes: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: definitely yes |  | 0
  Cycle 29 Day 15: probably yes: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15: probably yes |  | 0

28. Secondary Outcome: Percentage of Participants With Response to 'Patient Experience and Satisfaction End of Treatment Questionnaire (PESQ-EOT)'
Description: The PESQ-EOT consisting of 17 items assessed participant experience and satisfaction regarding the injection method (discomfort, pain, side effects, time saving and satisfaction) and study medication (side effects, worth taking, satisfaction and recommendation) and has been adapted based on qualitative interviews with oncology participants. In addition to the above, this questionnaire also includes additional items to assess whether participants received oncology medications in the past 2 years and if a participant received both IV and SC in the past 2 years, then participant preference on injection method (whether SC or IV). Percentage of participants with response to these additional items (received oncology medications in the past 2 years via IV/SC/both and if received both IV and SC; then the participant preference on injection method) are reported here. Percentages are rounded off to the tenth decimal place.
Time Frame: EOT visit (30 days after last study medication administration or before further anti myeloma therapy initiation, whichever occurred first, up to approximately 28 months)
Population: The ITT population included all randomized population. Only those participants with data collected at EOT are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 70 | 78
percentage of participants
  Received oncology medications in the past 2 years via IV only | 58.6 | 32.1
  Received oncology medications in the past 2 years via SC only | 12.9 | 23.1
  Received oncology medications in the past 2 years via both IV and SC | 12.9 | 20.5
  If received via both IV and SC: Preference for injection method: IV: number analyzed (Participants) | 9 | 16
  If received via both IV and SC: Preference for injection method: IV | 11.1 | 0
  If received via both IV and SC: Preference for injection method: SC: number analyzed (Participants) | 9 | 16
  If received via both IV and SC: Preference for injection method: SC | 33.3 | 87.5
  If received via both IV and SC: No preference for injection method: number analyzed (Participants) | 9 | 16
  If received via both IV and SC: No preference for injection method | 55.6 | 12.5

29. Secondary Outcome: Participant Responses to Patient's Assessment of Treatment (PAT) Questionnaire
Description: The 4-item PAT is an internally developed non-disease specific and self-administered assessment which has been debriefed with oncology patients during qualitative interviews. It provided participant insights on the benefits and disadvantages of treatment. Benefits and disadvantages were respectively rated on a 0-10 scale wherein 0=none (not beneficial at all or no disadvantages at all) and 10=maximum (extremely beneficial or extremely disadvantageous). Disadvantages vs benefits were rated on a scale of -3 to 3 wherein -3=disadvantages significantly outweigh the benefits, 0=equal benefits and disadvantages and 3=benefits significantly outweigh the disadvantages. Mean of benefits, disadvantages and disadvantages vs benefits is presented here.
Time Frame: as for outcome 28
Population: The ITT population included all randomized population. Only those participants with data collected at EOT for this endpoint are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 70 | 77
score on a scale
  Benefits | 5.7 (2.5) | 6.4 (2.3)
  Disadvantages | 4.3 (2.6) | 3.7 (2.6)
  Disadvantages vs benefits | 0.5 (2.0) | 1.2 (1.8)

30. Secondary Outcome: Health Resource Utilization and Productivity Questionnaire (HRUPQ): Baseline Healthcare Utilization: Number of Times in the Past 6 Months a Participant Received Care
Description: Healthcare utilization at baseline before study medication administration was collected via HRUPQ. The mean number of times in the past 6 months a participant received care in a clinic or hospital emergency room for any health issue including MM or due to MM and at-home care from a nurse or other health professional for any health issue including MM or due to MM is presented. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: Baseline (Cycle 1 Day 1)
Population: The ITT population included all randomized population. Only those participants with responses at Baseline are presented.
Measure: Mean (Standard Deviation); unit: number of times received care
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 51 | 74
number of times received care
  In a clinic or hospital emergency room for any health issue including MM | 3.6 (3.6) | 3.7 (4.1)
  In a clinic or hospital emergency room due to MM: number analyzed (Participants) | 47 | 52
  In a clinic or hospital emergency room due to MM | 4.4 (3.3) | 4.2 (4.2)
  At-home from nurse or other health professional for any health issue including MM: number analyzed (Participants) | 14 | 26
  At-home from nurse or other health professional for any health issue including MM | 4.4 (5.4) | 3.8 (3.2)
  At-home from nurse or other health professional due to MM: number analyzed (Participants) | 12 | 19
  At-home from nurse or other health professional due to MM | 4.7 (5.9) | 3.9 (3.6)

31. Secondary Outcome: HRUPQ: Baseline Healthcare Utilization: Number of Nights in the Past 6 Months a Participant Stayed in Hospital
Description: Healthcare utilization at baseline before study medication administration was collected via HRUPQ. The mean number of nights in the past 6 month a participant stayed in hospital for any health issue including MM or due to MM and stayed in intensive care unit (ICU) for any health issue including MM or due to MM is presented. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: Baseline (Cycle 1 Day 1)
Population: The ITT population included all randomized population. Only those participants with responses at Baseline are presented.
Measure: Mean (Standard Deviation); unit: number of nights
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 50 | 62
number of nights
  Stayed in hospital for any health issue including MM | 7.2 (12.3) | 5.2 (9.0)
  Stayed in hospital due to MM: number analyzed (Participants) | 38 | 37
  Stayed in hospital due to MM | 10.3 (20.2) | 6.5 (10.3)
  Stayed in ICU for any health issue including MM: number analyzed (Participants) | 3 | 6
  Stayed in ICU for any health issue including MM | 5.0 (2.6) | 1.3 (0.5)
  Stayed in ICU due to MM: number analyzed (Participants) | 0 | 3
  Stayed in ICU due to MM |  | 3.0 (2.0)

32. Secondary Outcome: HRUPQ: Baseline Healthcare Utilization: Number of Times in the Past 6 Months a Participant Consulted a Healthcare Professional (HCP)
Description: Healthcare utilization at baseline before study medication administration was collected via HRUPQ. The mean number of times in the past 6 months a participant consulted (had seen or talked to) following healthcare professionals: general doctor or primary care clinician (PCC) who treats a variety of illnesses for any health issue including MM or related to MM, physical or occupational therapist for any health issue including MM or related to MM, mental health professional (e.g. psychiatrist, psychologist, psychiatric nurse) for any health issue including MM or related to MM, medical doctor or clinician who specializes in particular medical disease or issue (specialist) for any health issue including MM or related to MM is presented. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: Baseline (Cycle 1 Day 1)
Population: The ITT population included all randomized population. Only those participants with responses at Baseline are presented.
Measure: Mean (Standard Deviation); unit: number of times consulted a HCP
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 113 | 110
number of times consulted a HCP
  General doctor or PCC for any health issue including MM | 4.5 (3.9) | 4.9 (5.4)
  General doctor or PCC for health issue related to MM: number analyzed (Participants) | 101 | 89
  General doctor or PCC for health issue related to MM | 4.5 (3.9) | 5.3 (7.6)
  Physical or occupational therapist for any health issue including MM: number analyzed (Participants) | 25 | 35
  Physical or occupational therapist for any health issue including MM | 6.3 (5.3) | 6.7 (9.7)
  Physical or occupational therapist for health issue related to MM: number analyzed (Participants) | 21 | 26
  Physical or occupational therapist for health issue related to MM | 6.2 (5.4) | 5.0 (6.4)
  Mental health professional for any health issue including MM: number analyzed (Participants) | 18 | 17
  Mental health professional for any health issue including MM | 3.2 (3.0) | 5.2 (7.4)
  Mental health professional for health issue related to MM: number analyzed (Participants) | 16 | 13
  Mental health professional for health issue related to MM | 3.3 (2.4) | 4.4 (7.8)
  Medical doctor or clinician (specialist) for any health issue including MM: number analyzed (Participants) | 76 | 80
  Medical doctor or clinician (specialist) for any health issue including MM | 4.2 (3.1) | 4.4 (3.3)
  Medical doctor or clinician (specialist) for health issue related to MM: number analyzed (Participants) | 77 | 79
  Medical doctor or clinician (specialist) for health issue related to MM | 4.5 (3.0) | 4.2 (2.4)

33. Secondary Outcome: Duration of Hospital Visits for Treatment Administration and Duration of Post-Treatment Monitoring Based on HRUPQ
Description: Medical resource utilization was collected through HRUPQ. Participants were asked to indicate the duration of their hospital visit (from arrival to departure) and the duration of post-treatment monitoring based on their most recent isatuximab administration. The median duration across all visits (starting from Cycle 2) was calculated and reported here.
Time Frame: From Cycle 2 Day 1 up to EOT visit (30 days after last study medication administration or before further anti myeloma therapy initiation, whichever occurred first, up to approximately 28 months)
Population: The ITT population included all randomized population.
Measure: Median (Full Range); unit: minutes
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 268 | 263
minutes
  Duration of hospital visit | 240.00 [1.0 to 500.0] | 180.00 [1.0 to 600.0]
  Duration of post-treatment monitoring | 30.00 [1.0 to 500.0] | 30.00 [1.0 to 500.0]

34. Secondary Outcome: Percentage of Participants Who Visited Healthcare Professional for Non-trial-related Health Issues Based on HRUPQ
Description: Medical resource utilization was collected through HRUPQ. Percentage of participants with healthcare professional visit not required by clinical trial since last isatuximab administration was recorded. Percentages are rounded off to the tenth decimal place.
Time Frame: Cycle 1 Days 8, 15 and 22, Cycle 2 Day 1, Cycles 3 to 29 Day 15 and EOT visit (30 days after last study medication administration or before further anti myeloma therapy initiation, whichever occurred first, up to approximately 28 months)
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 224 | 208
percentage of participants
  Cycle 1 Day 8: number analyzed (Participants) | 210 | 208
  Cycle 1 Day 8 | 11.4 | 14.9
  Cycle 1 Day 15: number analyzed (Participants) | 201 | 195
  Cycle 1 Day 15 | 10.0 | 9.2
  Cycle 1 Day 22: number analyzed (Participants) | 206 | 193
  Cycle 1 Day 22 | 11.7 | 9.8
  Cycle 2 Day 1: number analyzed (Participants) | 224 | 204
  Cycle 2 Day 1 | 12.5 | 10.8
  Cycle 3 Day 15: number analyzed (Participants) | 190 | 182
  Cycle 3 Day 15 | 13.2 | 11.5
  Cycle 4 Day 15: number analyzed (Participants) | 175 | 176
  Cycle 4 Day 15 | 13.1 | 8.5
  Cycle 5 Day 15: number analyzed (Participants) | 192 | 178
  Cycle 5 Day 15 | 8.9 | 7.3
  Cycle 6 Day 15: number analyzed (Participants) | 165 | 163
  Cycle 6 Day 15 | 9.7 | 9.2
  Cycle 7 Day 15: number analyzed (Participants) | 151 | 141
  Cycle 7 Day 15 | 13.2 | 9.2
  Cycle 8 Day 15: number analyzed (Participants) | 132 | 123
  Cycle 8 Day 15 | 16.7 | 14.6
  Cycle 9 Day 15: number analyzed (Participants) | 112 | 99
  Cycle 9 Day 15 | 11.6 | 14.1
  Cycle 10 Day 15: number analyzed (Participants) | 92 | 92
  Cycle 10 Day 15 | 10.9 | 14.1
  Cycle 11 Day 15: number analyzed (Participants) | 92 | 77
  Cycle 11 Day 15 | 13.0 | 10.4
  Cycle 12 Day 15: number analyzed (Participants) | 73 | 64
  Cycle 12 Day 15 | 6.8 | 10.9
  Cycle 13 Day 15: number analyzed (Participants) | 65 | 57
  Cycle 13 Day 15 | 16.9 | 12.3
  Cycle 14 Day 15: number analyzed (Participants) | 56 | 52
  Cycle 14 Day 15 | 12.5 | 5.8
  Cycle 15 Day 15: number analyzed (Participants) | 48 | 48
  Cycle 15 Day 15 | 18.8 | 12.5
  Cycle 16 Day 15: number analyzed (Participants) | 40 | 36
  Cycle 16 Day 15 | 7.5 | 13.9
  Cycle 17 Day 15: number analyzed (Participants) | 33 | 30
  Cycle 17 Day 15 | 15.2 | 16.7
  Cycle 18 Day 15: number analyzed (Participants) | 23 | 25
  Cycle 18 Day 15 | 13.0 | 12.0
  Cycle 19 Day 15: number analyzed (Participants) | 24 | 22
  Cycle 19 Day 15 | 8.3 | 13.6
  Cycle 20 Day 15: number analyzed (Participants) | 16 | 19
  Cycle 20 Day 15 | 12.5 | 15.8
  Cycle 21 Day 15: number analyzed (Participants) | 12 | 10
  Cycle 21 Day 15 | 25.0 | 0
  Cycle 22 Day 15: number analyzed (Participants) | 9 | 9
  Cycle 22 Day 15 | 44.4 | 11.1
  Cycle 23 Day 15: number analyzed (Participants) | 4 | 9
  Cycle 23 Day 15 | 0 | 22.2
  Cycle 24 Day 15: number analyzed (Participants) | 5 | 4
  Cycle 24 Day 15 | 20.0 | 0
  Cycle 25 Day 15: number analyzed (Participants) | 3 | 4
  Cycle 25 Day 15 | 0 | 25.0
  Cycle 26 Day 15: number analyzed (Participants) | 2 | 4
  Cycle 26 Day 15 | 0 | 0
  Cycle 27 Day 15: number analyzed (Participants) | 1 | 3
  Cycle 27 Day 15 | 0 | 0
  Cycle 28 Day 15: number analyzed (Participants) | 0 | 2
  Cycle 28 Day 15 |  | 50.0
  Cycle 29 Day 15: number analyzed (Participants) | 0 | 1
  Cycle 29 Day 15 |  | 0
  EOT visit: number analyzed (Participants) | 68 | 76
  EOT visit | 25.0 | 17.1

35. Secondary Outcome: Percentage of Participants Who Ever Retired During the Study Based on HRUPQ
Description: Employment status was assessed via HRUPQ. Percentage of participants who ever retired during the study are reported. Percentages are rounded off to the tenth decimal place.
Time Frame: From first dose of study medication administration (Day 1) up to PCD (06-Nov-2024), approximately 28 months
Population: The ITT population included all randomized population. Only those participants with data collected are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 252 | 250
percentage of participants | 81.7 | 83.6

36. Secondary Outcome: Percentage of Participants Who Retired Early Due to MM Based on HRUPQ
Description: Employment status was assessed via HRUPQ. Percentage of participants who retired early due to MM are reported. Percentages are rounded off to the tenth decimal place.
Time Frame: From first dose of study medication administration (Day 1) up to PCD (06-Nov-2024), approximately 28 months
Population: The ITT population included all randomized population. Only participants who retired during the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 206 | 209
percentage of participants | 32.0 | 37.3

37. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30): Global Health Status (GHS)/Quality of Life (QoL)
Description: EORTC QLQ-C30 is a cancer specific 30-item instrument that provides a comprehensive assessment of the principal health related QoL dimensions: GHS/QoL (2 items), functional scales (physical [5 items], role [2 items], emotional [4 items], cognitive [2 items], social [2 items]), symptom scales (fatigue [3 items], nausea & vomiting [2 items], pain [2 items]) and symptom items- 1 item each (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). For GHS/QoL: overall health and quality of life were assessed, rated on a 7-point scale (1: very poor to 7: excellent). All of the scales and single-item measures range in score from 0 to 100; mean is presented here. A higher score for GHS/QoL and a positive change from baseline represents a healthy/better level of QoL. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: Baseline (Cycle 1 Day 1) and Cycle 2 Day 1, Cycles 3 to 21 Day 15 and EOT visit (30 days after last study medication administration or before further anti myeloma therapy initiation, whichever occurred first, up to approximately 28 months)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 197
score on a scale
  Cycle 2 Day 1 | -2.78 (18.61) | -1.52 (17.79)
  Cycle 3 Day 15: number analyzed (Participants) | 165 | 175
  Cycle 3 Day 15 | -0.56 (19.15) | -0.52 (17.92)
  Cycle 4 Day 15: number analyzed (Participants) | 156 | 170
  Cycle 4 Day 15 | -0.05 (19.16) | 1.08 (19.20)
  Cycle 5 Day 15: number analyzed (Participants) | 166 | 161
  Cycle 5 Day 15 | 0.65 (18.49) | 1.04 (20.45)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | 0.34 (18.13) | 2.80 (19.56)
  Cycle 7 Day 15: number analyzed (Participants) | 131 | 130
  Cycle 7 Day 15 | -0.06 (20.56) | 2.24 (20.27)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 109
  Cycle 8 Day 15 | 2.85 (17.06) | -0.61 (20.56)
  Cycle 9 Day 15: number analyzed (Participants) | 100 | 84
  Cycle 9 Day 15 | 1.42 (20.55) | -0.99 (20.39)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 80
  Cycle 10 Day 15 | 2.34 (19.21) | 2.60 (19.24)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 68
  Cycle 11 Day 15 | 0.41 (18.70) | -0.86 (21.56)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 51
  Cycle 12 Day 15 | 2.56 (19.37) | 0.65 (23.85)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 45
  Cycle 13 Day 15 | 3.16 (19.17) | 6.11 (19.41)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 43
  Cycle 14 Day 15 | 4.33 (19.07) | 0.19 (22.75)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 15 | 1.70 (20.46) | 0.83 (22.86)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 31
  Cycle 16 Day 15 | 4.06 (16.87) | 2.42 (26.54)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 25
  Cycle 17 Day 15 | 3.33 (17.73) | 0.00 (25.00)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 20
  Cycle 18 Day 15 | 4.58 (17.20) | 2.08 (25.20)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 17
  Cycle 19 Day 15 | 2.65 (20.80) | -6.37 (20.74)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 14
  Cycle 20 Day 15 | 0.60 (12.43) | 0.60 (18.62)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | -3.33 (26.12) | 3.13 (16.63)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | -6.72 (22.42) | -4.11 (24.06)

38. Secondary Outcome: Change From Baseline in EORTC QLQ-C30: Physical Functioning
Description: EORTC QLQ-C30 is a cancer specific 30-item instrument that provides a comprehensive assessment of the principal health related QoL dimensions: GHS/QoL (2 items), functional scales (physical [5 items], role [2 items], emotional [4 items], cognitive [2 items], social [2 items]), symptom scales (fatigue [3 items], nausea & vomiting [2 items], pain [2 items]) and symptom items- 1 item each (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). For functional scales: questions were rated on a 4-point scale (1: not at all to 4: very much). All of the scales and single-item measures range in score from 0 to 100; mean is presented here. A higher score and a positive change from baseline represents a better level of physical functioning. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 197
score on a scale
  Cycle 2 Day 1 | -1.62 (17.20) | -2.10 (15.32)
  Cycle 3 Day 15: number analyzed (Participants) | 165 | 175
  Cycle 3 Day 15 | -1.98 (15.74) | -0.88 (16.96)
  Cycle 4 Day 15: number analyzed (Participants) | 156 | 170
  Cycle 4 Day 15 | -0.98 (14.62) | -1.33 (18.67)
  Cycle 5 Day 15: number analyzed (Participants) | 166 | 161
  Cycle 5 Day 15 | -1.41 (15.23) | -0.62 (18.15)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | -1.10 (14.82) | 0.37 (17.50)
  Cycle 7 Day 15: number analyzed (Participants) | 131 | 130
  Cycle 7 Day 15 | -2.04 (15.60) | -1.64 (17.63)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 109
  Cycle 8 Day 15 | -1.02 (15.68) | -0.55 (19.82)
  Cycle 9 Day 15: number analyzed (Participants) | 100 | 84
  Cycle 9 Day 15 | -1.93 (16.80) | -2.62 (17.35)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 80
  Cycle 10 Day 15 | -0.81 (15.16) | -0.92 (19.17)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 68
  Cycle 11 Day 15 | -2.20 (13.94) | -2.45 (17.31)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 51
  Cycle 12 Day 15 | -0.51 (12.60) | -1.96 (18.39)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 45
  Cycle 13 Day 15 | 0.11 (14.27) | -4.00 (19.46)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 43
  Cycle 14 Day 15 | 1.07 (12.22) | -4.50 (18.73)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 15 | -1.97 (17.70) | -2.33 (23.12)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 31
  Cycle 16 Day 15 | -0.17 (18.89) | -4.30 (21.74)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 25
  Cycle 17 Day 15 | -2.22 (16.36) | -4.00 (25.24)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 20
  Cycle 18 Day 15 | -3.00 (17.77) | -0.33 (22.21)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 17
  Cycle 19 Day 15 | -3.33 (19.27) | -7.84 (11.84)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 14
  Cycle 20 Day 15 | 0.48 (10.28) | -8.10 (14.83)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | -6.67 (16.33) | -2.50 (15.09)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | -7.96 (21.45) | -8.83 (20.71)

39. Secondary Outcome: Change From Baseline in EORTC QLQ-C30: Role Functioning
Description: EORTC QLQ-C30 is a cancer specific 30-item instrument that provides a comprehensive assessment of the principal health related QoL dimensions: GHS/QoL (2 items), functional scales (physical [5 items], role [2 items], emotional [4 items], cognitive [2 items], social [2 items]), symptom scales (fatigue [3 items], nausea & vomiting [2 items], pain [2 items]) and symptom items- 1 item each (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). For functional scales: questions were rated on a 4-point scale (1: not at all to 4: very much). All of the scales and single-item measures range in score from 0 to 100; mean is presented here. A higher score and a positive change from baseline represents a better level of role functioning. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 197
score on a scale
  Cycle 2 Day 1 | -4.59 (22.67) | -1.35 (24.24)
  Cycle 3 Day 15: number analyzed (Participants) | 165 | 175
  Cycle 3 Day 15 | -2.42 (22.86) | -1.24 (26.68)
  Cycle 4 Day 15: number analyzed (Participants) | 156 | 170
  Cycle 4 Day 15 | -0.75 (22.43) | 1.57 (26.48)
  Cycle 5 Day 15: number analyzed (Participants) | 166 | 161
  Cycle 5 Day 15 | -2.71 (20.70) | -0.62 (28.56)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | -1.84 (21.79) | -0.57 (27.43)
  Cycle 7 Day 15: number analyzed (Participants) | 131 | 130
  Cycle 7 Day 15 | -3.56 (23.48) | 0.00 (28.30)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 109
  Cycle 8 Day 15 | -1.35 (20.98) | -5.50 (32.24)
  Cycle 9 Day 15: number analyzed (Participants) | 100 | 84
  Cycle 9 Day 15 | -2.67 (20.20) | -6.55 (29.27)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 80
  Cycle 10 Day 15 | -2.85 (17.92) | -1.25 (27.40)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 68
  Cycle 11 Day 15 | -2.44 (17.98) | -8.33 (30.13)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 51
  Cycle 12 Day 15 | -1.79 (17.95) | -5.88 (28.64)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 45
  Cycle 13 Day 15 | -1.15 (17.06) | -4.07 (26.15)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 43
  Cycle 14 Day 15 | -2.33 (16.50) | -7.36 (33.79)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 15 | -3.03 (18.07) | -12.08 (32.68)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 31
  Cycle 16 Day 15 | -2.99 (17.88) | -10.22 (33.52)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 25
  Cycle 17 Day 15 | -3.89 (12.13) | -12.00 (37.74)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 20
  Cycle 18 Day 15 | -3.33 (15.86) | -3.33 (26.27)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 17
  Cycle 19 Day 15 | -3.03 (11.07) | -9.80 (19.60)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 14
  Cycle 20 Day 15 | -3.57 (9.65) | -13.10 (22.81)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | -11.67 (20.86) | 2.08 (27.37)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | -9.14 (25.90) | -8.92 (26.70)

40. Secondary Outcome: Change From Baseline in EORTC QLQ-C30: Emotional Functioning
Description: EORTC QLQ-C30 is a cancer specific 30-item instrument that provides a comprehensive assessment of the principal health related QoL dimensions: GHS/QoL (2 items), functional scales (physical [5 items], role [2 items], emotional [4 items], cognitive [2 items], social [2 items]), symptom scales (fatigue [3 items], nausea & vomiting [2 items], pain [2 items]) and symptom items- 1 item each (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). For functional scales: questions were rated on a 4-point scale (1: not at all to 4: very much). All of the scales and single-item measures range in score from 0 to 100; mean is presented here. A higher score and a positive change from baseline represents a better level of emotional functioning. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 197
score on a scale
  Cycle 2 Day 1 | -1.37 (17.91) | 2.28 (17.85)
  Cycle 3 Day 15: number analyzed (Participants) | 165 | 175
  Cycle 3 Day 15 | 0.71 (14.50) | 1.10 (19.02)
  Cycle 4 Day 15: number analyzed (Participants) | 156 | 170
  Cycle 4 Day 15 | -0.27 (17.52) | 3.14 (19.98)
  Cycle 5 Day 15: number analyzed (Participants) | 166 | 161
  Cycle 5 Day 15 | 0.35 (17.39) | 1.50 (18.14)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | 1.84 (17.28) | 1.37 (19.00)
  Cycle 7 Day 15: number analyzed (Participants) | 131 | 130
  Cycle 7 Day 15 | 0.64 (19.57) | 0.58 (20.81)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 109
  Cycle 8 Day 15 | 2.18 (18.21) | 1.07 (19.38)
  Cycle 9 Day 15: number analyzed (Participants) | 100 | 84
  Cycle 9 Day 15 | 0.33 (18.72) | 1.59 (23.48)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 80
  Cycle 10 Day 15 | 1.32 (17.78) | 3.44 (19.96)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 68
  Cycle 11 Day 15 | 0.10 (18.63) | 3.31 (23.88)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 51
  Cycle 12 Day 15 | 1.92 (18.79) | 4.74 (23.29)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 45
  Cycle 13 Day 15 | 3.02 (18.71) | -0.37 (23.16)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 43
  Cycle 14 Day 15 | 6.00 (19.49) | -0.78 (22.70)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 15 | 3.22 (19.87) | -0.21 (23.30)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 31
  Cycle 16 Day 15 | 3.85 (16.98) | -0.54 (22.46)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 25
  Cycle 17 Day 15 | 1.11 (15.43) | -1.33 (27.18)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 20
  Cycle 18 Day 15 | 4.58 (14.68) | -1.67 (19.79)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 17
  Cycle 19 Day 15 | 3.03 (17.36) | -7.84 (20.30)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 14
  Cycle 20 Day 15 | 2.38 (21.29) | -6.55 (18.25)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | 3.33 (16.29) | 3.13 (15.39)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | -5.24 (18.31) | -2.93 (20.42)

41. Secondary Outcome: Change From Baseline in EORTC QLQ-C30: Cognitive Functioning
Description: EORTC QLQ-C30 is a cancer specific 30-item instrument that provides a comprehensive assessment of the principal health related QoL dimensions: GHS/QoL (2 items), functional scales (physical [5 items], role [2 items], emotional [4 items], cognitive [2 items], social [2 items]), symptom scales (fatigue [3 items], nausea & vomiting [2 items], pain [2 items]) and symptom items- 1 item each (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). For functional scales: questions were rated on a 4-point scale (1: not at all to 4: very much). All of the scales and single-item measures range in score from 0 to 100; mean is presented here. A higher score and a positive change from baseline represents a better level of cognitive functioning. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 197
score on a scale
  Cycle 2 Day 1 | -1.32 (16.03) | 0.08 (19.53)
  Cycle 3 Day 15: number analyzed (Participants) | 165 | 175
  Cycle 3 Day 15 | -1.21 (18.37) | -2.00 (19.43)
  Cycle 4 Day 15: number analyzed (Participants) | 156 | 170
  Cycle 4 Day 15 | -1.07 (18.71) | 0.88 (17.70)
  Cycle 5 Day 15: number analyzed (Participants) | 166 | 161
  Cycle 5 Day 15 | -2.51 (16.68) | 0.00 (18.91)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | -2.30 (16.85) | -0.23 (17.62)
  Cycle 7 Day 15: number analyzed (Participants) | 131 | 130
  Cycle 7 Day 15 | -1.78 (17.69) | -1.03 (18.65)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 109
  Cycle 8 Day 15 | -2.40 (15.55) | -1.99 (20.75)
  Cycle 9 Day 15: number analyzed (Participants) | 100 | 84
  Cycle 9 Day 15 | -3.50 (17.13) | 1.39 (17.59)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 80
  Cycle 10 Day 15 | -4.47 (16.37) | -0.42 (19.84)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 68
  Cycle 11 Day 15 | -5.89 (18.21) | 0.49 (19.94)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 51
  Cycle 12 Day 15 | -4.62 (18.28) | 3.27 (21.35)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 45
  Cycle 13 Day 15 | -4.02 (16.90) | 0.74 (20.09)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 43
  Cycle 14 Day 15 | -4.00 (20.64) | -2.71 (21.19)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 15 | -6.44 (24.17) | -1.25 (19.75)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 31
  Cycle 16 Day 15 | -3.42 (21.69) | -3.76 (17.06)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 25
  Cycle 17 Day 15 | -2.78 (16.43) | -6.67 (22.05)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 20
  Cycle 18 Day 15 | -9.17 (17.50) | -5.00 (12.21)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 17
  Cycle 19 Day 15 | -6.82 (15.99) | -11.76 (15.33)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 14
  Cycle 20 Day 15 | -8.33 (16.98) | -13.10 (16.25)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | -18.33 (18.34) | -4.17 (14.77)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | -8.33 (24.66) | -0.23 (26.50)

42. Secondary Outcome: Change From Baseline in EORTC QLQ-C30: Social Functioning
Description: EORTC QLQ-C30 is a cancer specific 30-item instrument that provides a comprehensive assessment of the principal health related QoL dimensions: GHS/QoL (2 items), functional scales (physical [5 items], role [2 items], emotional [4 items], cognitive [2 items], social [2 items]), symptom scales (fatigue [3 items], nausea & vomiting [2 items], pain [2 items]) and symptom items- 1 item each (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). For functional scales: questions were rated on a 4-point scale (1: not at all to 4: very much). All of the scales and single-item measures range in score from 0 to 100; mean is presented here. A higher score and a positive change from baseline represents a better level of social functioning. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 197
score on a scale
  Cycle 2 Day 1 | -0.88 (21.66) | 0.17 (21.23)
  Cycle 3 Day 15: number analyzed (Participants) | 165 | 175
  Cycle 3 Day 15 | -0.51 (21.73) | 2.38 (24.35)
  Cycle 4 Day 15: number analyzed (Participants) | 156 | 170
  Cycle 4 Day 15 | -0.11 (20.08) | 2.06 (25.01)
  Cycle 5 Day 15: number analyzed (Participants) | 166 | 161
  Cycle 5 Day 15 | 0.40 (22.69) | 1.24 (23.98)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | -0.92 (24.75) | 1.48 (23.81)
  Cycle 7 Day 15: number analyzed (Participants) | 131 | 130
  Cycle 7 Day 15 | 1.53 (23.15) | 2.82 (25.43)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 109
  Cycle 8 Day 15 | 0.75 (23.50) | 0.76 (24.89)
  Cycle 9 Day 15: number analyzed (Participants) | 100 | 84
  Cycle 9 Day 15 | 3.67 (24.46) | -0.79 (22.98)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 80
  Cycle 10 Day 15 | 0.61 (24.07) | 0.21 (21.30)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 68
  Cycle 11 Day 15 | -0.61 (23.05) | 2.45 (25.31)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 51
  Cycle 12 Day 15 | 4.10 (24.30) | 0.65 (24.94)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 45
  Cycle 13 Day 15 | 2.30 (21.73) | 3.33 (22.08)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 43
  Cycle 14 Day 15 | 3.33 (19.05) | -2.33 (22.59)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 15 | 4.17 (20.69) | 1.25 (27.58)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 31
  Cycle 16 Day 15 | 4.27 (20.49) | -1.08 (22.33)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 25
  Cycle 17 Day 15 | 6.11 (22.09) | 5.33 (25.33)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 20
  Cycle 18 Day 15 | 7.50 (16.64) | -2.50 (18.16)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 17
  Cycle 19 Day 15 | 8.33 (18.37) | -0.98 (25.32)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 14
  Cycle 20 Day 15 | 8.33 (23.34) | -3.57 (22.81)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | 6.67 (22.50) | 18.75 (28.78)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | -4.84 (22.26) | -4.93 (32.90)

43. Secondary Outcome: Change From Baseline in EORTC QLQ-C30: Fatigue
Description: EORTC QLQ-C30 is a cancer specific 30-item instrument that provides a comprehensive assessment of the principal health related QoL dimensions: GHS/QoL (2 items), functional scales (physical [5 items], role [2 items], emotional [4 items], cognitive [2 items], social [2 items]), symptom scales (fatigue [3 items], nausea & vomiting [2 items], pain [2 items]) and symptom items- 1 item each (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). For symptom scales: questions were rated on a 4-point scale (1: not at all to 4: very much). All of the scales and single-item measures range in score from 0 to 100; mean is presented here. A higher score for symptoms and a positive change from baseline represents a higher level of symptomatology. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 197
score on a scale
  Cycle 2 Day 1 | 3.64 (20.33) | 4.00 (19.91)
  Cycle 3 Day 15: number analyzed (Participants) | 165 | 175
  Cycle 3 Day 15 | 3.91 (21.49) | 2.41 (20.28)
  Cycle 4 Day 15: number analyzed (Participants) | 156 | 170
  Cycle 4 Day 15 | 0.71 (19.70) | 1.18 (20.16)
  Cycle 5 Day 15: number analyzed (Participants) | 166 | 161
  Cycle 5 Day 15 | 1.41 (19.04) | 0.97 (20.62)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | -0.92 (20.05) | 0.53 (20.85)
  Cycle 7 Day 15: number analyzed (Participants) | 131 | 130
  Cycle 7 Day 15 | 0.93 (18.80) | 0.77 (20.90)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 109
  Cycle 8 Day 15 | 0.10 (18.98) | 2.85 (24.45)
  Cycle 9 Day 15: number analyzed (Participants) | 100 | 84
  Cycle 9 Day 15 | 1.89 (22.11) | 2.25 (21.11)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 80
  Cycle 10 Day 15 | -0.41 (22.12) | 1.39 (20.49)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 68
  Cycle 11 Day 15 | 2.30 (20.49) | 2.61 (19.40)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 51
  Cycle 12 Day 15 | 0.17 (17.29) | -1.09 (19.28)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 45
  Cycle 13 Day 15 | -3.07 (19.72) | 2.22 (19.04)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 43
  Cycle 14 Day 15 | -3.33 (18.54) | 3.62 (20.39)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 15 | 0.00 (20.47) | 2.78 (21.61)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 31
  Cycle 16 Day 15 | 1.42 (23.94) | 5.02 (21.44)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 25
  Cycle 17 Day 15 | 3.70 (20.91) | -0.44 (25.56)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 20
  Cycle 18 Day 15 | 1.67 (17.01) | -1.67 (16.63)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 17
  Cycle 19 Day 15 | 8.08 (18.84) | 3.92 (18.40)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 14
  Cycle 20 Day 15 | 11.90 (18.21) | 5.56 (17.84)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | 14.44 (26.22) | -6.94 (25.15)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | 7.89 (26.18) | 3.44 (22.89)

44. Secondary Outcome: Change From Baseline in EORTC QLQ-C30: Nausea and Vomiting
Description: as for outcome 43
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 197
score on a scale
  Cycle 2 Day 1 | 0.44 (13.14) | 1.18 (12.31)
  Cycle 3 Day 15: number analyzed (Participants) | 165 | 175
  Cycle 3 Day 15 | -2.22 (10.34) | -0.67 (13.29)
  Cycle 4 Day 15: number analyzed (Participants) | 156 | 170
  Cycle 4 Day 15 | -1.92 (11.19) | 0.49 (14.09)
  Cycle 5 Day 15: number analyzed (Participants) | 166 | 161
  Cycle 5 Day 15 | -1.20 (11.97) | 0.00 (13.31)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | -2.76 (11.62) | 0.57 (10.43)
  Cycle 7 Day 15: number analyzed (Participants) | 131 | 130
  Cycle 7 Day 15 | -1.27 (11.06) | -0.26 (12.45)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 109
  Cycle 8 Day 15 | -0.90 (11.42) | -0.46 (14.07)
  Cycle 9 Day 15: number analyzed (Participants) | 100 | 84
  Cycle 9 Day 15 | 0.33 (14.41) | -0.79 (11.25)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 80
  Cycle 10 Day 15 | 0.41 (11.70) | -0.21 (14.16)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 68
  Cycle 11 Day 15 | -1.63 (16.06) | 0.25 (13.66)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 51
  Cycle 12 Day 15 | -1.03 (14.70) | 1.31 (11.95)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 45
  Cycle 13 Day 15 | -2.87 (14.35) | 0.74 (16.27)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 43
  Cycle 14 Day 15 | -1.67 (17.90) | 3.10 (15.96)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 15 | -1.14 (15.42) | -0.83 (12.49)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 31
  Cycle 16 Day 15 | -2.14 (12.20) | 1.08 (15.48)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 25
  Cycle 17 Day 15 | 1.11 (12.33) | 1.33 (19.20)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 20
  Cycle 18 Day 15 | 0.83 (12.65) | 0.00 (5.41)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 17
  Cycle 19 Day 15 | 0.76 (19.57) | 1.96 (10.00)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 14
  Cycle 20 Day 15 | -2.38 (12.84) | 1.19 (10.26)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | 1.67 (18.34) | -2.08 (13.91)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | 2.96 (22.69) | -2.35 (16.74)

45. Secondary Outcome: Change From Baseline in EORTC QLQ-C30: Pain
Description: as for outcome 43
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 197
score on a scale
  Cycle 2 Day 1 | -3.79 (26.72) | -5.84 (24.48)
  Cycle 3 Day 15: number analyzed (Participants) | 165 | 175
  Cycle 3 Day 15 | -6.36 (22.50) | -8.76 (25.88)
  Cycle 4 Day 15: number analyzed (Participants) | 156 | 170
  Cycle 4 Day 15 | -7.48 (19.70) | -6.57 (25.21)
  Cycle 5 Day 15: number analyzed (Participants) | 166 | 161
  Cycle 5 Day 15 | -6.22 (21.82) | -8.70 (26.09)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | -6.90 (21.57) | -8.22 (26.42)
  Cycle 7 Day 15: number analyzed (Participants) | 131 | 130
  Cycle 7 Day 15 | -6.49 (22.98) | -8.46 (28.70)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 109
  Cycle 8 Day 15 | -7.51 (20.19) | -2.75 (26.21)
  Cycle 9 Day 15: number analyzed (Participants) | 100 | 84
  Cycle 9 Day 15 | -11.00 (23.83) | -3.17 (26.82)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 80
  Cycle 10 Day 15 | -7.32 (22.24) | -6.67 (28.39)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 68
  Cycle 11 Day 15 | -6.30 (22.78) | -7.60 (26.30)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 51
  Cycle 12 Day 15 | -6.41 (24.06) | -7.52 (27.14)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 45
  Cycle 13 Day 15 | -6.03 (22.01) | -5.93 (28.24)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 43
  Cycle 14 Day 15 | -9.00 (19.11) | -1.16 (31.37)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 15 | -3.79 (19.64) | -3.33 (29.77)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 31
  Cycle 16 Day 15 | -4.70 (22.28) | -4.30 (29.18)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 25
  Cycle 17 Day 15 | -1.67 (21.15) | -3.33 (37.58)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 20
  Cycle 18 Day 15 | -4.17 (20.14) | -2.50 (28.24)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 17
  Cycle 19 Day 15 | 0.00 (23.57) | -0.98 (25.32)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 14
  Cycle 20 Day 15 | -1.19 (20.11) | 1.19 (28.09)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | 6.67 (22.50) | -12.50 (24.80)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | -0.81 (33.26) | 4.69 (23.43)

46. Secondary Outcome: Change From Baseline in EORTC QLQ-C30: Dyspnea
Description: EORTC QLQ-C30 is a cancer specific 30-item instrument that provides a comprehensive assessment of the principal health related QoL dimensions: GHS/QoL (2 items), functional scales (physical [5 items], role [2 items], emotional [4 items], cognitive [2 items], social [2 items]), symptom scales (fatigue [3 items], nausea & vomiting [2 items], pain [2 items]) and symptom items- 1 item each (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). For symptom items: questions were rated on a 4-point scale (1: not at all to 4: very much). All of the scales and single-item measures range in score from 0 to 100; mean is presented here. A higher score for symptom items and a positive change from baseline represents a higher level of symptomatology. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 197
score on a scale
  Cycle 2 Day 1 | 5.11 (22.35) | 3.72 (21.50)
  Cycle 3 Day 15: number analyzed (Participants) | 165 | 175
  Cycle 3 Day 15 | 6.87 (25.10) | 1.33 (22.13)
  Cycle 4 Day 15: number analyzed (Participants) | 156 | 170
  Cycle 4 Day 15 | 4.91 (22.97) | 1.96 (20.09)
  Cycle 5 Day 15: number analyzed (Participants) | 166 | 161
  Cycle 5 Day 15 | 3.01 (24.84) | 3.73 (21.41)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | 4.60 (23.77) | 3.20 (19.70)
  Cycle 7 Day 15: number analyzed (Participants) | 131 | 130
  Cycle 7 Day 15 | 5.09 (24.28) | 3.08 (19.22)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 109
  Cycle 8 Day 15 | 7.81 (25.80) | 5.81 (21.20)
  Cycle 9 Day 15: number analyzed (Participants) | 100 | 84
  Cycle 9 Day 15 | 7.33 (24.88) | 4.76 (20.79)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 80
  Cycle 10 Day 15 | 5.28 (17.74) | 3.33 (19.56)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 68
  Cycle 11 Day 15 | 8.13 (22.57) | 4.41 (19.02)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 51
  Cycle 12 Day 15 | 6.67 (22.20) | 6.54 (24.96)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 45
  Cycle 13 Day 15 | 7.47 (23.40) | 8.15 (22.65)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 43
  Cycle 14 Day 15 | 6.00 (23.99) | 5.43 (22.92)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 15 | 9.85 (22.25) | 8.33 (23.57)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 31
  Cycle 16 Day 15 | 5.98 (24.03) | 7.53 (22.29)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 25
  Cycle 17 Day 15 | 10.00 (17.83) | 6.67 (21.52)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 20
  Cycle 18 Day 15 | 6.67 (23.20) | 8.33 (23.88)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 17
  Cycle 19 Day 15 | 7.58 (22.84) | 17.65 (31.44)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 14
  Cycle 20 Day 15 | 4.76 (25.68) | 4.76 (17.82)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | 16.67 (36.00) | 0.00 (17.82)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | 9.14 (26.43) | 4.23 (21.77)

47. Secondary Outcome: Change From Baseline in EORTC QLQ-C30: Insomnia
Description: as for outcome 46
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 197
score on a scale
  Cycle 2 Day 1 | 0.71 (27.71) | -3.89 (27.39)
  Cycle 3 Day 15: number analyzed (Participants) | 165 | 175
  Cycle 3 Day 15 | -4.24 (26.84) | -4.57 (29.33)
  Cycle 4 Day 15: number analyzed (Participants) | 156 | 170
  Cycle 4 Day 15 | -5.34 (25.54) | -8.04 (30.24)
  Cycle 5 Day 15: number analyzed (Participants) | 166 | 161
  Cycle 5 Day 15 | -4.62 (29.11) | -2.90 (30.14)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | -3.68 (27.81) | -4.57 (28.40)
  Cycle 7 Day 15: number analyzed (Participants) | 131 | 130
  Cycle 7 Day 15 | -1.27 (26.60) | -0.51 (30.50)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 109
  Cycle 8 Day 15 | -1.20 (27.31) | -6.12 (27.65)
  Cycle 9 Day 15: number analyzed (Participants) | 100 | 84
  Cycle 9 Day 15 | -2.33 (28.53) | -5.16 (31.26)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 80
  Cycle 10 Day 15 | -0.81 (24.55) | -4.58 (30.35)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 68
  Cycle 11 Day 15 | 2.03 (27.89) | -0.98 (26.99)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 51
  Cycle 12 Day 15 | -1.54 (27.28) | -3.27 (26.04)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 45
  Cycle 13 Day 15 | -5.17 (27.78) | -7.41 (25.51)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 43
  Cycle 14 Day 15 | -2.67 (30.00) | -3.88 (26.44)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 15 | 5.30 (32.90) | -5.83 (22.50)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 31
  Cycle 16 Day 15 | 0.85 (31.98) | 0.00 (25.82)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 25
  Cycle 17 Day 15 | -2.22 (27.59) | -2.67 (30.31)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 20
  Cycle 18 Day 15 | -3.33 (26.27) | -1.67 (27.52)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 17
  Cycle 19 Day 15 | -4.55 (25.81) | 5.88 (26.97)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 14
  Cycle 20 Day 15 | -2.38 (24.33) | 4.76 (25.68)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | 0.00 (22.22) | 0.00 (30.86)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | -5.91 (31.67) | -4.23 (32.82)

48. Secondary Outcome: Change From Baseline in EORTC QLQ-C30: Appetite Loss
Description: as for outcome 46
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 197
score on a scale
  Cycle 2 Day 1 | -0.18 (22.67) | 1.35 (20.71)
  Cycle 3 Day 15: number analyzed (Participants) | 165 | 175
  Cycle 3 Day 15 | -4.44 (18.60) | -2.48 (23.71)
  Cycle 4 Day 15: number analyzed (Participants) | 156 | 170
  Cycle 4 Day 15 | -4.06 (21.86) | -0.39 (22.64)
  Cycle 5 Day 15: number analyzed (Participants) | 166 | 161
  Cycle 5 Day 15 | -3.41 (20.64) | -0.83 (24.14)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | -6.44 (22.67) | -3.42 (23.07)
  Cycle 7 Day 15: number analyzed (Participants) | 131 | 130
  Cycle 7 Day 15 | -5.60 (20.74) | -1.79 (21.29)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 109
  Cycle 8 Day 15 | -4.80 (20.02) | -1.83 (23.93)
  Cycle 9 Day 15: number analyzed (Participants) | 100 | 84
  Cycle 9 Day 15 | -3.33 (28.62) | -1.98 (21.55)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 80
  Cycle 10 Day 15 | -3.66 (20.96) | -1.67 (23.66)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 68
  Cycle 11 Day 15 | -1.22 (26.94) | -1.47 (24.73)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 51
  Cycle 12 Day 15 | -3.08 (27.46) | -1.31 (22.07)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 45
  Cycle 13 Day 15 | -1.15 (22.48) | -5.19 (23.52)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 43
  Cycle 14 Day 15 | -1.33 (32.96) | -3.10 (22.79)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 15 | -3.03 (25.74) | -1.67 (27.16)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 31
  Cycle 16 Day 15 | -8.55 (26.18) | -2.15 (30.95)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 25
  Cycle 17 Day 15 | -5.56 (17.69) | -2.67 (27.08)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 20
  Cycle 18 Day 15 | -5.00 (22.36) | 0.00 (15.29)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 17
  Cycle 19 Day 15 | -3.03 (25.01) | 3.92 (11.07)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 14
  Cycle 20 Day 15 | -4.76 (22.10) | 7.14 (23.31)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | -3.33 (24.60) | 0.00 (0.00)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | 6.99 (36.78) | 3.76 (30.63)

49. Secondary Outcome: Change From Baseline in EORTC QLQ-C30: Constipation
Description: as for outcome 46
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 197
score on a scale
  Cycle 2 Day 1 | 4.76 (25.63) | 3.89 (27.80)
  Cycle 3 Day 15: number analyzed (Participants) | 165 | 175
  Cycle 3 Day 15 | 5.86 (26.79) | 9.52 (29.00)
  Cycle 4 Day 15: number analyzed (Participants) | 156 | 170
  Cycle 4 Day 15 | 6.41 (24.57) | 8.04 (28.68)
  Cycle 5 Day 15: number analyzed (Participants) | 166 | 161
  Cycle 5 Day 15 | 7.23 (27.97) | 5.59 (29.16)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | 6.90 (23.54) | 5.71 (29.13)
  Cycle 7 Day 15: number analyzed (Participants) | 131 | 130
  Cycle 7 Day 15 | 7.12 (26.80) | 4.62 (30.15)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 109
  Cycle 8 Day 15 | 6.91 (28.11) | 0.92 (27.39)
  Cycle 9 Day 15: number analyzed (Participants) | 100 | 84
  Cycle 9 Day 15 | 4.67 (26.39) | 1.98 (22.17)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 80
  Cycle 10 Day 15 | 2.44 (23.88) | 6.25 (27.61)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 68
  Cycle 11 Day 15 | 4.07 (20.55) | 5.39 (26.77)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 51
  Cycle 12 Day 15 | 3.08 (17.40) | 1.96 (27.82)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 45
  Cycle 13 Day 15 | 5.75 (17.81) | 5.93 (26.86)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 43
  Cycle 14 Day 15 | 5.33 (19.47) | 10.08 (27.73)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 15 | 3.03 (20.10) | 2.50 (26.57)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 31
  Cycle 16 Day 15 | 1.71 (15.20) | 4.30 (31.90)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 25
  Cycle 17 Day 15 | 3.33 (20.25) | 14.67 (36.11)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 20
  Cycle 18 Day 15 | 3.33 (28.41) | 3.33 (37.31)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 17
  Cycle 19 Day 15 | 6.06 (24.42) | 1.96 (32.21)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 14
  Cycle 20 Day 15 | 9.52 (15.63) | 7.14 (26.73)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | 3.33 (18.92) | 12.50 (17.25)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | -0.54 (31.65) | 1.88 (27.54)

50. Secondary Outcome: Change From Baseline in EORTC QLQ-C30: Diarrhea
Description: as for outcome 46
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 197
score on a scale
  Cycle 2 Day 1 | -3.17 (21.78) | -3.38 (23.81)
  Cycle 3 Day 15: number analyzed (Participants) | 165 | 175
  Cycle 3 Day 15 | -4.65 (24.11) | -5.33 (23.37)
  Cycle 4 Day 15: number analyzed (Participants) | 156 | 170
  Cycle 4 Day 15 | -4.70 (19.84) | -2.16 (24.90)
  Cycle 5 Day 15: number analyzed (Participants) | 166 | 161
  Cycle 5 Day 15 | -4.22 (20.49) | -3.11 (23.51)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | -0.92 (21.13) | -3.42 (24.36)
  Cycle 7 Day 15: number analyzed (Participants) | 131 | 130
  Cycle 7 Day 15 | -2.54 (20.93) | -3.33 (27.17)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 109
  Cycle 8 Day 15 | -6.01 (21.18) | -5.50 (25.06)
  Cycle 9 Day 15: number analyzed (Participants) | 100 | 84
  Cycle 9 Day 15 | -3.67 (25.02) | -4.76 (26.46)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 80
  Cycle 10 Day 15 | 0.00 (27.22) | -2.92 (28.16)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 68
  Cycle 11 Day 15 | -2.85 (23.54) | -6.37 (25.92)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 51
  Cycle 12 Day 15 | -6.67 (22.20) | -7.84 (24.57)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 45
  Cycle 13 Day 15 | -2.30 (21.50) | -2.22 (28.78)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 43
  Cycle 14 Day 15 | -2.00 (19.53) | -5.43 (25.12)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 15 | -3.79 (22.98) | -2.50 (21.86)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 31
  Cycle 16 Day 15 | -5.13 (21.00) | -3.23 (17.96)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 25
  Cycle 17 Day 15 | -6.67 (18.36) | -1.33 (15.15)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 20
  Cycle 18 Day 15 | -5.00 (22.36) | -8.33 (14.81)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 17
  Cycle 19 Day 15 | -7.58 (25.05) | 5.88 (24.25)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 14
  Cycle 20 Day 15 | -2.38 (27.62) | -2.38 (27.62)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | -10.00 (31.62) | -8.33 (15.43)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | -1.08 (24.86) | -3.76 (24.91)

51. Secondary Outcome: Change From Baseline in EORTC QLQ-C30: Financial Difficulties
Description: EORTC QLQ-C30 is a cancer specific 30-item instrument that provides a comprehensive assessment of the principal health related QoL dimensions: GHS/QoL (2 items), functional scales (physical [5 items], role [2 items], emotional [4 items], cognitive [2 items], social [2 items]), symptom scales (fatigue [3 items], nausea & vomiting [2 items], pain [2 items]) and symptom items- 1 item each (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). For symptom items: questions were rated on a 4-point scale (1: not at all to 4: very much). All of the scales and single-item measures range in score from 0 to 100; mean is presented here. A higher score for symptom items and a positive change from baseline represents a higher level of financial difficulties. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 189 | 197
score on a scale
  Cycle 2 Day 1 | -2.82 (21.56) | -5.08 (24.45)
  Cycle 3 Day 15: number analyzed (Participants) | 165 | 175
  Cycle 3 Day 15 | -2.63 (22.69) | -4.38 (28.59)
  Cycle 4 Day 15: number analyzed (Participants) | 156 | 170
  Cycle 4 Day 15 | -1.50 (22.51) | -3.33 (27.77)
  Cycle 5 Day 15: number analyzed (Participants) | 166 | 161
  Cycle 5 Day 15 | -3.61 (22.33) | -3.73 (29.81)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | -0.92 (21.13) | -3.42 (31.25)
  Cycle 7 Day 15: number analyzed (Participants) | 131 | 130
  Cycle 7 Day 15 | -2.04 (23.66) | -5.13 (30.06)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 109
  Cycle 8 Day 15 | -3.90 (21.90) | -4.59 (32.86)
  Cycle 9 Day 15: number analyzed (Participants) | 100 | 84
  Cycle 9 Day 15 | -2.67 (23.06) | -5.56 (29.65)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 80
  Cycle 10 Day 15 | -5.28 (22.51) | -7.50 (29.99)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 68
  Cycle 11 Day 15 | -2.85 (20.42) | -9.80 (30.51)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 51
  Cycle 12 Day 15 | -3.59 (23.66) | -3.92 (32.42)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 45
  Cycle 13 Day 15 | -5.75 (23.48) | -6.67 (31.46)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 43
  Cycle 14 Day 15 | -5.33 (24.61) | -5.43 (26.16)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 40
  Cycle 15 Day 15 | -0.76 (30.06) | -7.50 (29.71)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 31
  Cycle 16 Day 15 | -5.98 (25.21) | 1.08 (26.50)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 25
  Cycle 17 Day 15 | -7.78 (18.94) | -10.67 (31.51)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 20
  Cycle 18 Day 15 | -8.33 (26.21) | 0.00 (28.61)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 17
  Cycle 19 Day 15 | -6.06 (24.42) | 0.00 (26.35)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 14
  Cycle 20 Day 15 | -7.14 (26.73) | 11.90 (24.83)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | -16.67 (23.57) | -4.17 (33.03)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | 1.61 (22.12) | -2.82 (36.40)

52. Secondary Outcome: Change From Baseline in EORTC QLQ-Myeloma Module (MY20): Disease Symptoms
Description: The EORTC QLQ-MY20 was used in conjunction with the EORTC QLQ-C30 to assess symptoms and side effects due to the treatment or the disease which impacts health related QoL in participants with MM. It contains 20 items, 4 independent subscales covering 2 functional domains: symptom scales which include disease symptoms (6 items) and side-effects of treatment (10 items) and function scale which include future perspective (3 items) and body image (1 item). Scores for each subscale are based on the 4-point Likert scale ranging from (1: not at all to 4: very much) and transformed from raw scores to linear scales ranging from 0 to 100; mean is presented here. A higher score for disease symptoms and a positive change from baseline represents more symptoms, worse QoL. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 186 | 190
score on a scale
  Cycle 2 Day 1 | -4.63 (15.79) | -5.38 (15.67)
  Cycle 3 Day 15: number analyzed (Participants) | 160 | 169
  Cycle 3 Day 15 | -5.28 (15.74) | -5.92 (17.82)
  Cycle 4 Day 15: number analyzed (Participants) | 152 | 160
  Cycle 4 Day 15 | -5.08 (13.89) | -6.56 (16.95)
  Cycle 5 Day 15: number analyzed (Participants) | 165 | 158
  Cycle 5 Day 15 | -5.59 (16.55) | -8.33 (17.96)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | -6.63 (15.93) | -8.14 (19.15)
  Cycle 7 Day 15: number analyzed (Participants) | 130 | 130
  Cycle 7 Day 15 | -5.94 (15.87) | -8.21 (17.87)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 107
  Cycle 8 Day 15 | -4.75 (14.21) | -7.06 (19.16)
  Cycle 9 Day 15: number analyzed (Participants) | 99 | 83
  Cycle 9 Day 15 | -6.90 (16.99) | -7.70 (19.49)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 78
  Cycle 10 Day 15 | -6.23 (15.21) | -7.76 (19.00)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 66
  Cycle 11 Day 15 | -4.81 (13.82) | -9.60 (19.91)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 50
  Cycle 12 Day 15 | -4.62 (18.26) | -10.22 (18.52)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 44
  Cycle 13 Day 15 | -5.75 (17.69) | -5.43 (16.79)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 42
  Cycle 14 Day 15 | -8.11 (14.69) | -6.22 (16.88)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 39
  Cycle 15 Day 15 | -4.55 (16.26) | -6.13 (17.51)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 30
  Cycle 16 Day 15 | -7.12 (16.76) | -6.85 (16.42)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 24
  Cycle 17 Day 15 | -4.63 (13.69) | -6.94 (19.12)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 19
  Cycle 18 Day 15 | -1.11 (11.48) | -8.19 (19.80)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 16
  Cycle 19 Day 15 | 0.00 (12.36) | -6.94 (13.38)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 13
  Cycle 20 Day 15 | -1.19 (13.29) | -7.26 (15.28)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | 1.67 (10.81) | -8.33 (12.94)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | 1.08 (22.76) | 5.40 (20.70)

53. Secondary Outcome: Change From Baseline in EORTC QLQ-MY20: Side Effects of Treatment
Description: The EORTC QLQ-MY20 was used in conjunction with the EORTC QLQ-C30 to assess symptoms and side effects due to the treatment or the disease which impacts health related QoL in participants with MM. It contains 20 items, 4 independent subscales covering 2 functional domains: symptom scales which include disease symptoms (6 items) and side-effects of treatment (10 items) and function scale which include future perspective (3 items) and body image (1 item). Scores for each subscale are based on the 4-point Likert scale ranging from (1: not at all to 4: very much) and transformed from raw scores to linear scales ranging from 0 to 100; mean is presented here. A higher score for side effects of treatment and a positive change from baseline represents more side effects, worse QoL. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 186 | 190
score on a scale
  Cycle 2 Day 1 | 2.05 (11.38) | 0.30 (12.29)
  Cycle 3 Day 15: number analyzed (Participants) | 160 | 169
  Cycle 3 Day 15 | 1.68 (11.26) | 0.55 (13.29)
  Cycle 4 Day 15: number analyzed (Participants) | 152 | 160
  Cycle 4 Day 15 | 2.21 (12.34) | 0.14 (14.86)
  Cycle 5 Day 15: number analyzed (Participants) | 165 | 158
  Cycle 5 Day 15 | 2.51 (12.18) | 1.75 (15.08)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | 1.14 (13.20) | -0.50 (13.22)
  Cycle 7 Day 15: number analyzed (Participants) | 130 | 130
  Cycle 7 Day 15 | 1.42 (12.96) | 0.83 (15.31)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 107
  Cycle 8 Day 15 | 1.02 (13.10) | 0.81 (15.10)
  Cycle 9 Day 15: number analyzed (Participants) | 99 | 83
  Cycle 9 Day 15 | 1.33 (13.88) | 0.17 (14.46)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 78
  Cycle 10 Day 15 | 3.01 (12.71) | 0.10 (14.14)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 66
  Cycle 11 Day 15 | 2.20 (14.29) | 0.00 (15.46)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 50
  Cycle 12 Day 15 | 0.59 (12.19) | -2.27 (13.41)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 44
  Cycle 13 Day 15 | 1.37 (13.43) | -0.93 (13.38)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 42
  Cycle 14 Day 15 | 1.27 (13.61) | 0.36 (14.86)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 39
  Cycle 15 Day 15 | 2.46 (12.43) | -0.37 (12.93)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 30
  Cycle 16 Day 15 | 2.77 (13.08) | -0.32 (14.67)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 24
  Cycle 17 Day 15 | 3.25 (12.11) | -2.39 (15.70)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 19
  Cycle 18 Day 15 | 1.17 (12.07) | -1.81 (13.08)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 16
  Cycle 19 Day 15 | 3.08 (15.21) | 2.55 (12.98)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 13
  Cycle 20 Day 15 | 4.60 (16.56) | 4.22 (21.45)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | 4.48 (18.29) | -8.84 (16.10)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | 2.55 (13.61) | -0.23 (13.97)

54. Secondary Outcome: Change From Baseline in EORTC QLQ-MY20: Future Perspective
Description: The EORTC QLQ-MY20 was used in conjunction with the EORTC QLQ-C30 to assess symptoms and side effects due to the treatment or the disease which impacts health related QoL in participants with MM. It contains 20 items, 4 independent subscales covering 2 functional domains: symptom scales which include disease symptoms (6 items) and side-effects of treatment (10 items) and function scale which include future perspective (3 items) and body image (1 item). Scores for each subscale are based on the 4-point Likert scale ranging from (1: not at all to 4: very much) and transformed from raw scores to linear scales ranging from 0 to 100; mean is presented here. A higher score for future perspectives and a positive change from baseline represents better outcomes, better QoL. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 186 | 190
score on a scale
  Cycle 2 Day 1 | 2.75 (19.17) | 5.15 (19.72)
  Cycle 3 Day 15: number analyzed (Participants) | 160 | 169
  Cycle 3 Day 15 | 3.96 (20.68) | 6.38 (22.14)
  Cycle 4 Day 15: number analyzed (Participants) | 152 | 160
  Cycle 4 Day 15 | 5.41 (22.33) | 9.65 (24.14)
  Cycle 5 Day 15: number analyzed (Participants) | 165 | 158
  Cycle 5 Day 15 | 4.44 (22.72) | 8.44 (22.27)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | 4.67 (21.74) | 7.99 (23.59)
  Cycle 7 Day 15: number analyzed (Participants) | 130 | 130
  Cycle 7 Day 15 | 4.96 (21.92) | 6.92 (24.56)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 107
  Cycle 8 Day 15 | 5.81 (20.04) | 5.40 (23.06)
  Cycle 9 Day 15: number analyzed (Participants) | 99 | 83
  Cycle 9 Day 15 | 5.84 (22.69) | 7.50 (25.15)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 78
  Cycle 10 Day 15 | 5.15 (18.41) | 6.41 (23.79)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 66
  Cycle 11 Day 15 | 4.47 (18.55) | 3.70 (24.76)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 50
  Cycle 12 Day 15 | 5.47 (17.14) | 1.11 (26.20)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 44
  Cycle 13 Day 15 | 6.13 (17.92) | 3.28 (21.51)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 42
  Cycle 14 Day 15 | 8.22 (22.20) | 1.06 (23.26)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 39
  Cycle 15 Day 15 | 3.28 (21.38) | 1.99 (28.14)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 30
  Cycle 16 Day 15 | 7.41 (15.99) | 1.48 (26.54)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 24
  Cycle 17 Day 15 | 6.30 (16.93) | -0.46 (27.89)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 19
  Cycle 18 Day 15 | 5.00 (15.49) | -1.75 (28.99)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 16
  Cycle 19 Day 15 | 3.03 (18.84) | -8.33 (23.48)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 13
  Cycle 20 Day 15 | 6.35 (19.84) | -9.40 (17.48)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | 7.78 (18.92) | -1.39 (15.07)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | -1.97 (23.68) | -2.66 (25.30)

55. Secondary Outcome: Change From Baseline in EORTC QLQ-MY20: Body Image
Description: The EORTC QLQ-MY20 was used in conjunction with the EORTC QLQ-C30 to assess symptoms and side effects due to the treatment or the disease which impacts health related QoL in participants with MM. It contains 20 items, 4 independent subscales covering 2 functional domains: symptom scales which include disease symptoms (6 items) and side-effects of treatment (10 items) and function scale which include future perspective (3 items) and body image (1 item). Scores for each subscale are based on the 4-point Likert scale ranging from (1: not at all to 4: very much) and transformed from raw scores to linear scales ranging from 0 to 100; mean is presented here. A higher score for body image and a positive change from baseline represents better outcomes, better QoL. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 186 | 190
score on a scale
  Cycle 2 Day 1 | 3.23 (25.26) | 2.63 (26.76)
  Cycle 3 Day 15: number analyzed (Participants) | 160 | 169
  Cycle 3 Day 15 | 1.88 (26.50) | 1.78 (23.64)
  Cycle 4 Day 15: number analyzed (Participants) | 152 | 160
  Cycle 4 Day 15 | 0.88 (24.25) | 4.79 (25.31)
  Cycle 5 Day 15: number analyzed (Participants) | 165 | 158
  Cycle 5 Day 15 | -0.61 (27.17) | 2.95 (25.06)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 146
  Cycle 6 Day 15 | -0.92 (25.74) | 5.94 (26.75)
  Cycle 7 Day 15: number analyzed (Participants) | 130 | 130
  Cycle 7 Day 15 | -2.31 (28.21) | 3.85 (26.13)
  Cycle 8 Day 15: number analyzed (Participants) | 111 | 107
  Cycle 8 Day 15 | -2.70 (27.39) | 3.74 (24.37)
  Cycle 9 Day 15: number analyzed (Participants) | 99 | 83
  Cycle 9 Day 15 | 2.02 (26.00) | 5.62 (25.41)
  Cycle 10 Day 15: number analyzed (Participants) | 82 | 78
  Cycle 10 Day 15 | 0.81 (26.70) | 6.41 (26.89)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 66
  Cycle 11 Day 15 | -5.69 (26.09) | 6.06 (23.32)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 50
  Cycle 12 Day 15 | -2.05 (26.27) | 5.33 (21.68)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 44
  Cycle 13 Day 15 | -4.02 (31.27) | 5.30 (23.78)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 42
  Cycle 14 Day 15 | 0.00 (30.12) | 3.17 (20.57)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 39
  Cycle 15 Day 15 | -3.03 (35.08) | 4.27 (23.17)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 30
  Cycle 16 Day 15 | -2.56 (35.36) | 1.11 (23.95)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 24
  Cycle 17 Day 15 | 5.56 (32.85) | -4.17 (24.70)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 19
  Cycle 18 Day 15 | 8.33 (26.21) | 1.75 (17.48)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 16
  Cycle 19 Day 15 | 9.09 (27.57) | -2.08 (19.12)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 13
  Cycle 20 Day 15 | 7.14 (29.75) | -10.26 (31.58)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | 6.67 (37.84) | 8.33 (15.43)
  EOT visit: number analyzed (Participants) | 62 | 71
  EOT visit | -3.76 (30.84) | 1.88 (27.54)

56. Secondary Outcome: Change From Baseline in European Quality of Life Group Measure With 5 Dimensions and 5 Levels Per Dimension (EQ-5D-5L): Visual Analogue Scale (VAS)
Description: The EQ-5D-5L is a standardized measure of health status that provides a simple, generic measure of health utility, and consists of 2 sections: descriptive and a VAS. The descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The VAS records the respondent's self-rated health on a 20-cm vertical scale ranging from 0: the worst health you can imagine to 100: the best health you can imagine. Change from baseline in VAS is reported here. A higher score in VAS and positive change from baseline represents a better level of QoL. The baseline value was defined as the last non-missing value collected on or before the start date of study medication.
Time Frame: as for outcome 37
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 186 | 189
score on a scale
  Cycle 2 Day 1 | 0.99 (17.62) | -0.39 (14.58)
  Cycle 3 Day 15: number analyzed (Participants) | 159 | 168
  Cycle 3 Day 15 | -0.52 (17.35) | -0.10 (16.28)
  Cycle 4 Day 15: number analyzed (Participants) | 151 | 160
  Cycle 4 Day 15 | 0.75 (18.66) | -0.24 (19.36)
  Cycle 5 Day 15: number analyzed (Participants) | 164 | 157
  Cycle 5 Day 15 | 0.09 (17.78) | 1.03 (19.20)
  Cycle 6 Day 15: number analyzed (Participants) | 145 | 145
  Cycle 6 Day 15 | 0.50 (19.54) | 2.39 (18.17)
  Cycle 7 Day 15: number analyzed (Participants) | 130 | 126
  Cycle 7 Day 15 | -1.55 (20.69) | 3.02 (18.01)
  Cycle 8 Day 15: number analyzed (Participants) | 110 | 105
  Cycle 8 Day 15 | 0.12 (17.97) | -0.14 (18.03)
  Cycle 9 Day 15: number analyzed (Participants) | 98 | 82
  Cycle 9 Day 15 | 0.87 (19.39) | 0.62 (16.07)
  Cycle 10 Day 15: number analyzed (Participants) | 81 | 77
  Cycle 10 Day 15 | 2.65 (15.86) | 2.38 (15.85)
  Cycle 11 Day 15: number analyzed (Participants) | 82 | 64
  Cycle 11 Day 15 | -0.51 (20.30) | -1.66 (17.53)
  Cycle 12 Day 15: number analyzed (Participants) | 65 | 49
  Cycle 12 Day 15 | 1.97 (20.67) | -0.51 (17.55)
  Cycle 13 Day 15: number analyzed (Participants) | 58 | 44
  Cycle 13 Day 15 | 2.83 (18.71) | 3.41 (15.74)
  Cycle 14 Day 15: number analyzed (Participants) | 50 | 42
  Cycle 14 Day 15 | 1.58 (18.62) | -0.83 (17.36)
  Cycle 15 Day 15: number analyzed (Participants) | 44 | 39
  Cycle 15 Day 15 | 2.41 (20.90) | -1.69 (17.75)
  Cycle 16 Day 15: number analyzed (Participants) | 39 | 29
  Cycle 16 Day 15 | 2.38 (20.48) | 0.72 (19.44)
  Cycle 17 Day 15: number analyzed (Participants) | 30 | 23
  Cycle 17 Day 15 | 2.90 (18.33) | -0.13 (17.38)
  Cycle 18 Day 15: number analyzed (Participants) | 20 | 19
  Cycle 18 Day 15 | 3.45 (15.70) | 0.53 (23.17)
  Cycle 19 Day 15: number analyzed (Participants) | 22 | 16
  Cycle 19 Day 15 | -0.05 (18.17) | -6.00 (15.16)
  Cycle 20 Day 15: number analyzed (Participants) | 14 | 13
  Cycle 20 Day 15 | -2.14 (12.24) | -2.92 (21.34)
  Cycle 21 Day 15: number analyzed (Participants) | 10 | 8
  Cycle 21 Day 15 | -5.20 (24.93) | 1.88 (9.19)
  EOT visit: number analyzed (Participants) | 61 | 70
  EOT visit | -4.25 (21.94) | -5.17 (17.11)

57. Secondary Outcome: ORR Based on at Least 1 Chromosomal Abnormality
Description: BM aspirate was collected for fluorescent in situ hybridization for analysis of del[17p], t[4;14], t[14;16]) and 1q21+. ORR was also evaluated based on IRC assessment by disease characteristics. ORR for participants with at least 1 chromosomal abnormality i.e. [del(17p)] or [1q21+ and t(4;14) or t(14;16)] is presented. Percentages are rounded off to the tenth decimal place.
Time Frame: From first dose of study medication administration (Day 1) up to PCD (06-Nov-2024), approximately 28 months
Population: The ITT population included all randomized population. Only participants with at least 1 chromosomal abnormality are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
Number analyzed (Participants) | 53 | 48
percentage of participants | 60.4 | 62.5

ADVERSE EVENTS:
Time Frame: Adverse events and deaths were collected from first dose of study medication administration (Day 1) up to 30 days after the last dose of study medication, approximately 28 months. Interim results are presented up to PCD of 06-Nov-2024.
Description: Adverse events were collected for safety population. All-cause mortality was collected for the randomized population.
Arm/Group | Isa-IV + Pd | Isa-SC + Pd
All-Cause Mortality (participants affected / at risk) | 49/268 | 50/263
Serious Adverse Events (participants affected / at risk) | 127/264 | 139/263
Other Adverse Events (participants affected / at risk) | 241/264 | 234/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isa-IV + Pd (N=264) | Isa-SC + Pd (N=263)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bullous Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 7 (7) | 6 (6)
Covid-19 Pneumonia (Infections and infestations) | 6 (6) | 6 (6)
Campylobacter Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 2 (2)
Coronavirus Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cryptococcal Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Cryptosporidiosis Infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus Chorioretinitis (Infections and infestations) | 1 (1) | 1 (1)
Dengue Fever (Infections and infestations) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea Infectious (Infections and infestations) | 0 (0) | 1 (1)
Disseminated Cryptococcosis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis Escherichia Coli (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Salmonella (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal Infection (Infections and infestations) | 1 (1) | 0 (0)
Haematological Infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infective Exacerbation Of Asthma (Infections and infestations) | 0 (0) | 1 (1)
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 5 (5) | 1 (1)
Listeria Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Liver Abscess (Infections and infestations) | 1 (1) | 0 (0)
Localised Infection (Infections and infestations) | 0 (0) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 2 (2) | 3 (4)
Lower Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 1 (1)
Ludwig Angina (Infections and infestations) | 0 (0) | 1 (1)
Meningitis Cryptococcal (Infections and infestations) | 1 (1) | 0 (0)
Meningitis Listeria (Infections and infestations) | 1 (1) | 0 (0)
Meningococcal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Metapneumovirus Infection (Infections and infestations) | 0 (0) | 2 (2)
Metapneumovirus Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Neutropenic Infection (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae Virus Infection (Infections and infestations) | 1 (1) | 1 (1)
Pertussis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Pneumonia (Infections and infestations) | 36 (42) | 38 (41)
Pneumonia Adenoviral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia Cytomegaloviral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Escherichia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Influenzal (Infections and infestations) | 4 (4) | 3 (3)
Pneumonia Legionella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Parainfluenzae Viral (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia Pneumococcal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia Viral (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Syncytial Virus Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 (0) | 2 (2)
Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2)
Respiratory Tract Infection Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection Viral (Infections and infestations) | 1 (1) | 2 (2)
Rhinovirus Infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Septic Shock (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Soft Tissue Infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal Bacteraemia (Infections and infestations) | 1 (2) | 1 (1)
Staphylococcal Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Fungal Infection (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (5) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 5 (7)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (2)
Wound Infection Staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leptomeningeal Myelomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma Cell Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 5 (5)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 (6) | 9 (9)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Adrenal Disorder (Endocrine disorders) | 0 (0) | 1 (1)
Hypercalcaemia Of Malignancy (Endocrine disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0)
Drug Abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Cluster Headache (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Putamen Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Spinal Cord Compression (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (2) | 0 (0)
Toxic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal Neuralgia (Nervous system disorders) | 0 (0) | 1 (2)
Vocal Cord Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Cataract Nuclear (Eye disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 4 (4) | 3 (3)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Diverticular Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis Fulminant (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Scar Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Haematoma Muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 6 (6)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 2 (2)
Disease Progression (General disorders) | 6 (6) | 4 (4)
General Physical Health Deterioration (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Sudden Death (General disorders) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 1 (1) | 1 (1)
Blood Potassium Decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil Count Decreased (Investigations) | 1 (1) | 2 (2)
Platelet Count Decreased (Investigations) | 9 (9) | 4 (4)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Intentional Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isa-IV + Pd (N=264) | Isa-SC + Pd (N=263)
Bronchitis (Infections and infestations) | 17 (18) | 18 (22)
Covid-19 (Infections and infestations) | 33 (35) | 27 (29)
Influenza (Infections and infestations) | 4 (4) | 15 (15)
Nasopharyngitis (Infections and infestations) | 17 (22) | 16 (18)
Pneumonia (Infections and infestations) | 23 (24) | 18 (20)
Upper Respiratory Tract Infection (Infections and infestations) | 59 (91) | 60 (107)
Urinary Tract Infection (Infections and infestations) | 17 (20) | 11 (12)
Neutropenia (Blood and lymphatic system disorders) | 80 (158) | 84 (170)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (22) | 15 (17)
Insomnia (Psychiatric disorders) | 39 (58) | 39 (44)
Dizziness (Nervous system disorders) | 14 (16) | 19 (21)
Headache (Nervous system disorders) | 15 (19) | 12 (13)
Peripheral Sensory Neuropathy (Nervous system disorders) | 18 (21) | 19 (20)
Tremor (Nervous system disorders) | 17 (17) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (25) | 20 (25)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 14 (14)
Abdominal Pain (Gastrointestinal disorders) | 6 (8) | 15 (20)
Constipation (Gastrointestinal disorders) | 33 (40) | 38 (42)
Diarrhoea (Gastrointestinal disorders) | 53 (81) | 50 (63)
Nausea (Gastrointestinal disorders) | 21 (27) | 18 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (17) | 12 (13)
Back Pain (Musculoskeletal and connective tissue disorders) | 22 (24) | 25 (27)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 25 (33) | 16 (18)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 14 (14) | 7 (9)
Asthenia (General disorders) | 20 (24) | 20 (23)
Fatigue (General disorders) | 37 (41) | 51 (57)
Influenza Like Illness (General disorders) | 14 (22) | 12 (17)
Oedema Peripheral (General disorders) | 31 (35) | 22 (26)
Pyrexia (General disorders) | 17 (22) | 16 (22)
Neutrophil Count Decreased (Investigations) | 41 (60) | 46 (65)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 63 (67) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT05405166/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT05405166/SAP_001.pdf